CLINICAL TRIAL: NCT03692078
Title: A Randomized, Controlled, Study to Evaluate Changes in Exposure to Harmful and Potentially Harmful Constituents in Adult Smokers Who Partially or Completely Switch to Oral Tobacco-derived Nicotine Products in a Clinical Setting.
Brief Title: A Study to Evaluate Changes in Smokers Using Oral Tobacco-derived Nicotine Products.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altria Client Services LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ALCS-RDS-18-04-VRV
Record Dates: First submitted 2018-09-21; First posted 2018-10-02 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- GROUP 1: Continue Smoking (No Intervention): Subjects will be asked to continue smoking their own brand (OB) cigarettes ad libitum for 7 days.
- GROUP 2: OTDN product 1 (Experimental): Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline cigarettes per day (CPD) and use at least 3 oral tobacco-derived nicotine (OTDN) product units per day for 7 days.
  Interventions: Other: OTDN product 1
- GROUP 3: OTDN product 2 (Experimental): Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 oral tobacco-derived nicotine (OTDN) product units per day for 7 days.
  Interventions: Other: OTDN product 2
- GROUP 4: OTDN product 1 (Experimental): Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine (OTDN) product, using at least 3 OTDN product units per day for 7 days.
  Interventions: Other: OTDN product 1
- GROUP 5: OTDN product 2 (Experimental): Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine (OTDN) product, using at least 3 OTDN product units per day for 7 days.
  Interventions: Other: OTDN product 2
- GROUP 6: Tobacco Cessation (Experimental): Subjects will completely stop all tobacco product usage for 7 days.
  Interventions: Other: Tobacco Cessation

INTERVENTIONS:
Other: OTDN product 1 — Oral tobacco-derived nicotine product
  Arms: GROUP 2: OTDN product 1; GROUP 4: OTDN product 1
Other: OTDN product 2 — Oral tobacco-derived nicotine product
  Arms: GROUP 3: OTDN product 2; GROUP 5: OTDN product 2
Other: Tobacco Cessation — Tobacco Cessation
  Arms: GROUP 6: Tobacco Cessation

SUMMARY:
The purpose of this study is to evaluate changes in exposure to selected harmful and potentially harmful constituents (HPHC) by measuring biomarkers in adult smokers who partially or completely switch from smoking cigarettes to oral tobacco-derived nicotine (OTDN) products compared to those who continue exclusive smoking cigarettes or stop using all tobacco products.

DETAILED DESCRIPTION:
This is an open label, randomized, 6 parallel-group clinical study evaluating changes in exposure to selected HPHCs, subjective effects, and product use behavior in adult smokers relative to continued smoking who are randomly assigned to continue smoking, partially or completely switch to oral tobacco-derived nicotine products, or stop using any tobacco products for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary consent to participate in this study documented on the signed informed consent form (ICF).
2. Healthy adult males and females 21 to 65 years of age, inclusive, at Screening
3. Smoking history of an average of at least 10 but no more than 30 factory manufactured combustible cigarettes daily for at least 1 year prior to Screening. Brief periods (i.e., up to 7 consecutive days) of non-smoking during the 3 months prior to Screening (e.g., due to illness or participation in a study where smoking was prohibited) will be permitted.
4. Positive urine cotinine (≥ 500 ng/mL) at Screening.
5. Willing to comply with the requirements of the study.
6. Willing to use all test products after product trial at Check in.
7. Willing and able to abstain from cigarettes from Day 1 through the End of the study.

Exclusion Criteria:

1. Use of any type of tobacco or nicotine containing products other than manufactured cigarettes (e.g., e vapor products, roll-your-own cigarettes, bidis, snuff, nicotine inhaler, pipe, cigar, chewing tobacco, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum) in the 7 days prior to Check in
2. Self-reported puffers (i.e., adult smokers who draw smoke from the cigarette into the mouth and throat but do not inhale).
3. Planning to quit smoking in the next 30 days (from Screening visit).
4. History or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, existing respiratory diseases, immunologic, psychiatric, lymphatic, or cardiovascular disease, or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
5. Clinically significant abnormal findings on the vital signs, physical examination, medical history, ECG, or clinical laboratory results, in the opinion of the Investigator.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will enroll healthy adult male and female (no more than 60% of either gender) self affirmed combustible cigarette smokers, 21-65 years of age
Enrollment: 231 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios D Karles, PhD, Study Director — Altria Client Services LLC
Locations (2):
- United States (2):
  - QPS Bio-Kinetic Clinical Applications, LLC, Springfield, Missouri
  - Inflamax - Hill Top Research, Neptune City, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were required to complete a test product tolerability trial and baseline assessment over the course of 3 days prior to randomization on Day 1 of the study. A total of 213 subjects were randomized to one of the six groups in this study.
Groups:
- Product Trial: Subjects were enrolled in the product trial period but discontinued from the study prior to randomization.
- GROUP 1: Continue Smoking: Subjects will be asked to continue smoking their OB cigarettes ad libitum for 7 days.
- GROUP 2: OTDN Product 1: Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 product units per day for 7 days.
  OTDN product 1: Oral tobacco-derived nicotine product
- GROUP 3: OTDN Product 2: Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 product units per day for 7 days.
  OTDN product 2: Oral tobacco-derived nicotine product
- GROUP 4: OTDN Product 1: Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine product, using at least 3 product units per day for 7 days.
  OTDN product 1: Oral tobacco-derived nicotine product
- GROUP 5: OTDN Product 2: Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine product, using at least 3 product units per day for 7 days.
  OTDN product 2: Oral tobacco-derived nicotine product
Period: Overall Study
Arm/Group | Product Trial | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Started | 18 | 40 | 42 | 41 | 30 | 30 | 30
Completed | 0 | 38 | 42 | 40 | 25 | 26 | 27
Not Completed | 18 | 2 | 0 | 1 | 5 | 4 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Enrollment Closed | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Failure To Meet Randomization Criteria | 13 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1 | 5 | 3 | 3

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Product Trial: All subjects who used a study product during the product trial period, including subjects who were discontinued from the study before randomization and subjects who were randomized to one of the six study groups.
- GROUP 1: Continue Smoking: Subjects will be asked to continue smoking their own brand of cigarettes ad libitum for 7 days.
- GROUP 2: OTDN Product 1: Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 product units per day for 7 days.
  OTDN product 1: Oral tobacco-derived nicotine product (VERVE® Discs)
- GROUP 3: OTDN Product 2: Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 product units per day for 7 days.
  OTDN product 2: Oral tobacco-derived nicotine product (VERVE® Chews)
- GROUP 4: OTDN Product 1: Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine product, using at least 3 product units per day for 7 days.
  OTDN product 1: Oral tobacco-derived nicotine product (VERVE® Discs)
- GROUP 5: OTDN Product 2: Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine product, using at least 3 product units per day for 7 days.
  OTDN product 2: Oral tobacco-derived nicotine product (VERVE® Chews)
- Total: Total of all reporting groups
Arm/Group | Product Trial | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation | Total
Number analyzed (Participants) | 18 | 40 | 42 | 41 | 30 | 30 | 30 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11.48) | 36.6 (11.07) | 39.8 (11.60) | 43.7 (12.29) | 38.3 (12.62) | 38.2 (13.09) | 41.5 (8.11) | 39.8 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 19 | 15 | 15 | 12 | 12 | 96
  Male | 8 | 27 | 23 | 26 | 15 | 18 | 18 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 4 | 3 | 4 | 1 | 2 | 19
  Not Hispanic or Latino | 17 | 36 | 38 | 38 | 26 | 29 | 28 | 212
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian and Black | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  American Indian, Black, White | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 5 | 13 | 14 | 14 | 8 | 12 | 14 | 80
  Black, White | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 12 | 27 | 26 | 22 | 22 | 18 | 16 | 143
  Asian, White | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight [Mean (Standard Deviation); unit: kg] | 78.46 (15.918) | 84.07 (15.491) | 84.81 (16.063) | 86.75 (19.738) | 83.84 (18.142) | 78.57 (15.467) | 86.82 (13.220) | 84.31 (16.614)
Height [Mean (Standard Deviation); unit: cm] | 168.6 (10.19) | 172.7 (7.69) | 171.7 (8.96) | 172.2 (9.36) | 170.4 (9.86) | 171.6 (8.32) | 171.3 (9.15) | 171.7 (8.82)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 27.656 (5.3195) | 28.130 (4.6162) | 28.679 (4.6677) | 29.134 (5.4869) | 28.847 (5.3881) | 26.670 (5.1232) | 29.693 (4.7754) | 28.547 (5.0294)
Highest Grade of School [Count of Participants; unit: Participants]
  Elementary School | 1 | 4 | 0 | 0 | 2 | 0 | 0 | 7
  Some High School | 2 | 3 | 4 | 5 | 5 | 6 | 2 | 27
  High School Graduate | 5 | 17 | 19 | 19 | 17 | 11 | 13 | 101
  1-3 Years College | 8 | 13 | 12 | 16 | 4 | 9 | 10 | 72
  4+ Years College | 2 | 1 | 4 | 0 | 1 | 4 | 4 | 16
  Postgraduate/Masters/Doctorate/Law/MD | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 6
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Do Not Wish to Answer | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Annual Income [Count of Participants; unit: Participants]
  Under $20,000 | 8 | 16 | 13 | 14 | 13 | 10 | 13 | 87
  $20,000 - $29,999 | 3 | 9 | 13 | 12 | 7 | 13 | 3 | 60
  $30,000 - $39,999 | 4 | 4 | 8 | 11 | 6 | 3 | 5 | 41
  $40,000 - $49,999 | 1 | 1 | 1 | 2 | 1 | 1 | 2 | 9
  $50,000 - $59,999 | 1 | 3 | 0 | 1 | 0 | 1 | 1 | 7
  $60,000 - $74,999 | 1 | 4 | 1 | 0 | 0 | 1 | 4 | 11
  $75,000 - $99,999 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 4
  $100,000 - $149,999 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Do Not Wish to Answer | 0 | 1 | 4 | 1 | 2 | 0 | 2 | 10
Daily Cigarette Use [Mean (Standard Deviation); unit: Cigarettes per day] — Data was collected from subject responses at screening reporting the number of cigarettes smoked per day (CPD).
  Cigarettes per day | 16.8 (5.92) | 16.8 (4.61) | 17.8 (6.02) | 18.4 (5.99) | 15.9 (3.53) | 16.7 (5.35) | 17.8 (5.90) | 17.3 (5.37)
Years Smoked [Mean (Standard Deviation); unit: years] — Data collected from subject tobacco use history.
  years | 19.4 (13.23) | 17.6 (11.33) | 18.9 (12.22) | 23.6 (13.68) | 21.7 (13.38) | 12.93 (12.93) | 22.2 (9.36) | 20.8 (12.32)
Fagerström Test for Cigarette Dependence [Mean (Standard Deviation); unit: points] — The Fagerström Test assesses an individual's dependence on nicotine. It consists of Yes/No and multiple choice questions where each response is assigned a value from 0 to 1 (for yes/no questions) or 0 to 3 (for multiple choice questions). Values are summed to yield a total score with a minimum score of 0 points and a maximum score of 10 points. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
  points | 5.2 (2.13) | 5.9 (1.76) | 5.4 (1.62) | 5.2 (1.87) | 5.4 (1.43) | 5.6 (1.28) | 5.6 (1.61) | 5.5 (1.62)
Cigarette Brand Style History Summary [Count of Participants; unit: Participants] — Data was collected on subjects' own brand of cigarettes. The categories refer to cigarette brand, flavor, style and size, respectively.
  Participants
    NEWPORT, MENTHOL, GREEN, 100mm (100s) | 4 | 9 | 12 | 16 | 8 | 8 | 8 | 65
    NEWPORT, MENTHOL, GREEN, 85mm (Kings) | 0 | 2 | 1 | 2 | 0 | 2 | 6 | 13
    PALL MALL, NON MENTHOL, RED, 100mm (100s) | 0 | 2 | 1 | 3 | 1 | 2 | 1 | 10
    MARLBORO, NON MENTHOL, GOLD, 85mm (Kings) | 0 | 2 | 3 | 1 | 0 | 2 | 1 | 9
    MARLBORO, NON MENTHOL, BLACK, 100mm (100s) | 1 | 1 | 1 | 1 | 3 | 2 | 0 | 9
    L&M, NON MENTHOL, RED, 85mm (Kings) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 5
    MARLBORO, NON MENTHOL, RED, 100mm (100s) | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 5
    MARLBORO, NON MENTHOL, RED, 85mm (Kings) | 2 | 0 | 1 | 1 | 2 | 1 | 0 | 7
    PALL MALL, NON MENTHOL, BLUE, 100mm (100s) | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 6
    CAMEL, MENTHOL, CRUSH SILVER, 85mm (Kings) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 4
    NATURAL AMERICAN SPIRIT, NON MENTHOL, YELLOW, 85mm (Kings) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 4
    CAMEL, MENTHOL, CRUSH, 85mm (Kings) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3
    L&M, MENTHOL, GREEN, 100mm (100s) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
    L&M, MENTHOL, GREEN, 85mm (Kings) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3
    PALL MALL, MENTHOL, GREEN, 100mm (100s) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
    PALL MALL, MENTHOL, GREEN, 85mm (Kings) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
    BERLEY, MENTHOL, GREEN, 100mm (100s) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
    CAMEL, NON MENTHOL, WIDES FILTERS, 85mm (Kings) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
    DECADE, NON MENTHOL, RED, 100mm (100s) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
    KOOL, MENTHOL, GREEN, 100mm (100s) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
    MARLBORO, MENTHOL, BLACK, 85mm (Kings) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
    MARLBORO, MENTHOL, GOLD, 85mm (Kings) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
    MARLBORO, MENTHOL, MIDNIGHT, 85mm (Kings) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
    MARLBORO, MENTHOL, SMOOTH, 85mm (Kings) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
    MARLBORO, NON MENTHOL, BLACK, 85mm (Kings) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
    MARLBORO, NON MENTHOL, RED SPECIAL SELECT, 85mm (Kings) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 3
    NEWPORT, NON MENTHOL, RED, 85mm (Kings) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
    PALL MALL, NON MENTHOL, RED, 85mm (Kings) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
    BERLEY, NON MENTHOL, GOLD, 85mm (Kings) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    CAMEL, MENTHOL, WIDES DARK GREEN, 85mm (Kings) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    CAMEL, NON MENTHOL, BLUE, 85mm (Kings) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 3
    CAMEL, NON MENTHOL, FILTERS, 85mm (Kings) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    CAMEL, NON MENTHOL, TURKISH BLEND GOLD, 85mm (Kings) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    CHEYENNE, MENTHOL, GREEN, 100mm (100s) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    CHEYENNE, MENTHOL, GREEN, 85mm (Kings) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    CHEYENNE, NON MENTHOL, RED, 100mm (100s) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    DECADE, MENTHOL, GREEN, 100mm (100s) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    EAGLE 20'S, MENTHOL, GOLD, 100mm (100s) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    EDGEFIELD, NON MENTHOL, RED, 100mm (100s) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    EXETER, MENTHOL, GREEN, 100mm (100s) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    EXETER, NON MENTHOL, KINGS (RED), 85mm (Kings) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    EXETER, NON MENTHOL, RED, 100mm (100s) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    L&M, MENTHOL, DARK GREEN (GOLD PACK), 100mm (100s) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    L&M, MENTHOL, DARK GREEN FILTER, 100mm (100s) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    L&M, MENTHOL, DARK GREEN, 85mm (Kings) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    L&M, NON MENTHOL, RED, 100mm (100s) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    L&M, NON MENTHOL, TURKISH BLEND GOLD, 85mm (Kings) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 3
    LIGGETT, NON MENTHOL, RED, 85mm (Kings) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    MARLBORO, MENTHOL, GOLD, 100mm (100s) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    MARLBORO, MENTHOL, GREEN, 100mm (100s) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    MARLBORO, MENTHOL, GREEN, 72mm | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    MARLBORO, MENTHOL, NXT, 85mm (Kings) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    MARLBORO, NON MENTHOL, BLEND NO 27, 85mm (Kings) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    MARLBORO, NON MENTHOL, RED, 72mm | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    MARLBORO, NON MENTHOL, SOUTHERN CUT, 85mm (Kings) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    MARLBORO, NON MENTHOL, SPECIAL BLEND GOLD, 100mm (100s) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    MARLBORO, NON MENTHOL, SPECIAL BLEND GOLD, 85mm (Kings) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    MARLBORO, NON MENTHOL, SPECIAL BLEND RED, 100mm (100s) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    MARLBORO, NON MENTHOL, SPECIAL BLEND RED, 85mm (Kings) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    MAVERICK, MENTHOL, GREEN, 100mm (100s) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
    NEWPORT, MENTHOL, BLUE, 85mm (Kings) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    NEWPORT, MENTHOL, GREEN, 72mm | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    NEWPORT, NON MENTHOL, GOLD, 100mm (100s) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    NEWPORT, NON MENTHOL, RED, 100mm (100s) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    PALL MALL, MENTHOL, BLACK, 100mm (100s) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    PALL MALL, MENTHOL, WHITE, 100mm (100s) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    PALL MALL, NON MENTHOL, BLUE, 85mm (Kings) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    PALL MALL, NON MENTHOL, RED FILTER, 100mm (100s) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    PYRAMID, NON MENTHOL, RED, 72mm | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    SIGNAL, NON MENTHOL, RED, 85mm (Kings) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    USA GOLD, NON MENTHOL, GOLD, 85mm (Kings) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    WINSTON, NON MENTHOL, GOLD, 85mm (Kings) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    WINSTON, NON MENTHOL, RED, 85mm (Kings) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    L&M, NON MENTHOL, RED FILTER, 85mm (Kings) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    MARLBORO, NON MENTHOL, RED SPECIAL SELECT, 100mm (100s) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    NATURAL AMERICAN SPIRIT, NON MENTHOL, TURQUOISE, 85mm (Kings) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Summary of Urine Total NNAL Amount Excreted and Absolute Change From Baseline (ng/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of urine total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) amount excreted (ng/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the lower limit of quantitation (LLOQ) (2.00 pg/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: Modified ITT (mITT): All randomized subjects who used at least one study product after randomization (except Group 6) and had a valid baseline and at least one post-baseline biomarker measure
Measure: Mean (Standard Deviation); unit: ng/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ng/24 hour
  Day -1 | 511.889 (273.0646) | 581.676 (317.8968) | 548.751 (259.9637) | 638.849 (309.2360) | 599.162 (387.2946) | 527.260 (208.6977)
  Day 5 | 487.095 (276.4866) | 378.601 (225.0280) | 412.952 (252.9450) | 189.353 (109.4009) | 234.376 (183.1248) | 169.303 (77.4737)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 476.074 (296.5802) | 389.094 (226.8891) | 394.254 (240.8056) | 167.289 (100.1691) | 176.869 (135.1699) | 146.405 (60.3849)
  Change from Baseline (Day 5) | -24.795 (86.2810) | -203.075 (210.6622) | -135.800 (143.0520) | -449.496 (257.2221) | -364.786 (235.7564) | -357.958 (169.8953)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -35.816 (85.0846) | -173.010 (172.5258) | -154.497 (120.7393) | -460.402 (263.3910) | -407.814 (259.3657) | -371.172 (162.2706)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 6.116, 95% CI 2-sided [5.976 to 6.255] — LSM calculated from the mixed model for repeated measures that includes study group, day, group by day interaction, and gender as fixed effects, log transformed baseline value as covariate, with a covariance matrix based on the AIC value
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 6.073, 95% CI 2-sided [5.963 to 6.183] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.736, 95% CI 2-sided [5.605 to 5.868] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.792, 95% CI 2-sided [5.687 to 5.897] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.835, 95% CI 2-sided [5.701 to 5.969] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.799, 95% CI 2-sided [5.694 to 5.904] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.881, 95% CI 2-sided [4.713 to 5.048] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.844, 95% CI 2-sided [4.711 to 4.977] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.185, 95% CI 2-sided [5.021 to 5.350] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.933, 95% CI 2-sided [4.801 to 5.066] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.014, 95% CI 2-sided [4.852 to 5.175] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.892, 95% CI 2-sided [4.763 to 5.020] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0013, Mixed Models Analysis; Mean Difference (Net) = -0.379, 95% CI 2-sided [-0.646 to -0.112] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0034, Mixed Models Analysis; Mean Difference (Net) = -0.281, 95% CI 2-sided [-0.496 to -0.065] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0354, Mixed Models Analysis; Mean Difference (Net) = -0.281, 95% CI 2-sided [-0.549 to -0.012] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0044, Mixed Models Analysis; Mean Difference (Net) = -0.274, 95% CI 2-sided [-0.489 to -0.059] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.235, 95% CI 2-sided [-1.539 to -0.930] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.229, 95% CI 2-sided [-1.475 to -0.983] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.930, 95% CI 2-sided [-1.230 to -0.630] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.140, 95% CI 2-sided [-1.383 to -0.896] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.723, 95% CI 2-sided [0.436 to 1.009] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.901, 95% CI 2-sided [0.667 to 1.134] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.821, 95% CI 2-sided [0.533 to 1.109] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.907, 95% CI 2-sided [.675 to 1.140] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = .8291, Mixed Models Analysis; Mean Difference (Net) = -0.133, 95% CI 2-sided [-0.453 to 0.188] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.9997, Mixed Models Analysis; Mean Difference (Net) = -0.048, 95% CI 2-sided [-0.308 to 0.213] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.5755, Mixed Models Analysis; Mean Difference (Net) = 0.172, 95% CI 2-sided [-0.145 to 0.488] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: NNAL amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.9999, Mixed Models Analysis; Mean Difference (Net) = 0.042, 95% CI 2-sided [-0.217 to 0.301] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Summary of Urine Total NNAL Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of urine total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (2.00 pg/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: Modified ITT: All randomized subjects who used at least one study product after randomization (except Group 6) and had a valid baseline and at least one post-baseline biomarker measure
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | -4.241 (22.0910) | -31.755 (28.5666) | -26.092 (23.2887) | -66.540 (18.5833) | -61.140 (14.0247) | -67.092 (11.7400)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -8.377 (20.0357) | -29.261 (20.2229) | -29.854 (17.7150) | -70.823 (13.8839) | -68.763 (16.4492) | -71.244 (8.1469)

3. Secondary Outcome: Summary of NNN Amount Excreted and Absolute Change From Baseline (ng/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of N-nitrosonornicotine (NNN) amount excreted (ng/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.500 pg/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ng/24 hour
  Day -1 | 17.153 (14.5452) | 25.737 (32.2433) | 20.254 (12.7633) | 37.567 (93.0133) | 21.096 (17.4601) | 20.271 (15.2179)
  Day 5 | 15.718 (12.1674) | 14.414 (23.0907) | 13.367 (20.6899) | 1.524 (1.8065) | 5.535 (23.7712) | 0.968 (0.7968)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 16.221 (11.7555) | 34.944 (142.4443) | 26.542 (94.8042) | 0.902 (1.3344) | 1.876 (3.8928) | 1.166 (1.5528)
  Change from Baseline (Day 5) | -1.434 (6.2770) | -11.324 (20.7146) | -6.888 (21.1344) | -36.042 (92.0468) | -15.562 (27.2973) | -19.303 (15.2298)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -0.932 (7.8298) | 9.323 (143.0700) | 6.288 (95.6402) | -37.431 (94.9572) | -18.669 (16.6816) | -19.532 (15.8782)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.629, 95% CI 2-sided [2.317 to 2.940] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.632, 95% CI 2-sided [2.321 to 2.943] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.006, 95% CI 2-sided [1.714 to 2.298] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.143, 95% CI 2-sided [1.847 to 2.440] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.987, 95% CI 2-sided [1.690 to 2.284] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.261, 95% CI 2-sided [1.964 to 2.559] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p = 0.1658, Mixed Models Analysis; Mean Difference (Net) = -0.263, 95% CI 2-sided [-0.635 to 0.109] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p = 0.0007, Mixed Models Analysis; Mean Difference (Net) = -0.659, 95% CI 2-sided [-1.036 to -0.282] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Non-Inferiority — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p = 0.1055, Mixed Models Analysis; Mean Difference (Net) = -0.302, 95% CI 2-sided [-0.667 to 0.064] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p = 0.2040, Mixed Models Analysis; Mean Difference (Net) = -0.243, 95% CI 2-sided [-0.617 to 0.132] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p = 0.1829, Mixed Models Analysis; Mean Difference (Net) = -0.244, 95% CI 2-sided [-0.603 to 0.116] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p = 0.1801, Mixed Models Analysis; Mean Difference (Net) = -0.248, 95% CI 2-sided [-0.612 to 0.115] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0391, Mixed Models Analysis; Mean Difference (Net) = -0.622, 95% CI 2-sided [-1.225 to -0.019] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.1864, Mixed Models Analysis; Mean Difference (Net) = -0.489, 95% CI 2-sided [-1.096 to 0.119] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0310, Mixed Models Analysis; Mean Difference (Net) = -0.642, 95% CI 2-sided [-1.246 to -0.037] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0310, Mixed Models Analysis; Mean Difference (Net) = -0.642, 95% CI 2-sided [-1.246 to -0.037] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.891, 95% CI 2-sided [-3.580 to -2.202] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.291, 95% CI 2-sided [-3.985 to -2.597] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.930, 95% CI 2-sided [-3.605 to -2.255] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.875, 95% CI 2-sided [-3.559 to -2.190] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.250, 95% CI 2-sided [1.604 to 2.896] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.391, 95% CI 2-sided [1.737 to 3.046] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.231, 95% CI 2-sided [1.582 to 2.879] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.509, 95% CI 2-sided [1.857 to 3.162] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -0.019, 95% CI 2-sided [-0.743 to 0.705] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.5639, Mixed Models Analysis; Mean Difference (Net) = -0.411, 95% CI 2-sided [-1.142 to 0.320] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -0.058, 95% CI 2-sided [-0.771 to 0.656] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: NNN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.006, 95% CI 2-sided [-0.721 to 0.732] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Summary of NNN Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of N-nitrosonornicotine (NNN) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.500 pg/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | 17.679 (135.9950) | -39.207 (55.1440) | -29.116 (121.2696) | -90.367 (14.4687) | -79.576 (68.3202) | -89.967 (21.7083)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 11.041 (67.8187) | 39.909 (533.3498) | 110.644 (699.0961) | -93.379 (11.0686) | -88.301 (16.9805) | -73.064 (101.7367)

5. Secondary Outcome: Summary of Nicotine Equivalents Amount Excreted and Absolute Change From Baseline (mg/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of nicotine equivalents amount excreted (mg/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) for each metabolite were set to one-half of the LLOQ for the calculation of nicotine equivalents. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void). Nicotine equivalents (mg/g creatinine) = nicotine equivalents (μg/mL) x 100 / creatinine (mg/dL)
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
mg/24 hour
  Day -1 | 16.887 (5.4959) | 17.497 (5.9794) | 17.904 (7.1881) | 15.991 (5.8914) | 15.752 (4.9830) | 16.279 (4.9702)
  Day 5 | 16.297 (5.4573) | 12.330 (4.0796) | 15.024 (5.5730) | 5.459 (6.7089) | 8.191 (5.9189) | 0.668 (0.3787)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 16.832 (5.8963) | 12.832 (4.1984) | 15.363 (6.1114) | 5.476 (7.3802) | 7.437 (5.1587) | 0.481 (0.2954)
  Change from Baseline (Day 5) | -0.590 (3.3816) | -5.167 (4.8936) | -2.880 (4.7547) | -10.532 (6.5032) | -7.561 (6.9238) | -15.611 (4.8231)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -0.055 (3.6896) | -4.429 (3.9681) | -2.541 (4.6321) | -10.571 (7.2563) | -8.555 (6.1938) | -15.580 (4.8301)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: NE amount excreted (mg/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.691, 95% CI 2-sided [2.519 to 2.863] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: NE amount excreted (mg/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.718, 95% CI 2-sided [2.546 to 2.890] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: NE amount excreted (mg/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.415, 95% CI 2-sided [2.252 to 2.577] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: NE amount excreted (mg/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.440, 95% CI 2-sided [2.276 to 2.603] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: NE amount excreted (mg/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.583, 95% CI 2-sided [2.417 to 2.748] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: NE amount excreted (mg/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.591, 95% CI 2-sided [2.426 to 2.757] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: NE amount excreted (mg/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.107, 95% CI 2-sided [0.901 to 1.314] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: NE amount excreted (mg/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.017, 95% CI 2-sided [0.810 to 1.225] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: NE amount excreted (mg/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.828, 95% CI 2-sided [1.624 to 2.031] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: NE amount excreted (mg/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.782, 95% CI 2-sided [1.577 to 1.988] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: NE amount excreted (mg/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.550, 95% CI 2-sided [-0.750 to -0.350] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: NE amount excreted (mg/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.850, 95% CI 2-sided [-1.051 to -0.650] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: NE amount excreted (mg/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.1608, Mixed Models Analysis; Mean Difference (Net) = -0.276, 95% CI 2-sided [-0.609 to 0.057] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: NE amount excreted (mg/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.1575, Mixed Models Analysis; Mean Difference (Net) = -0.278, 95% CI 2-sided [-0.613 to 0.056] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: NE amount excreted (mg/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.9728, Mixed Models Analysis; Mean Difference (Net) = -0.108, 95% CI 2-sided [-0.442 to 0.226] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: NE amount excreted (mg/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.9262, Mixed Models Analysis; Mean Difference (Net) = -0.127, 95% CI 2-sided [-0.461 to 0.208] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: NE amount excreted (mg/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.584, 95% CI 2-sided [-1.963 to -1.204] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: NE amount excreted (mg/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.701, 95% CI 2-sided [-2.081 to -1.320] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: NE amount excreted (mg/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.863, 95% CI 2-sided [-1.237 to -0.489] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: NE amount excreted (mg/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: NE amount excreted (mg/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: NE amount excreted (mg/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.936, 95% CI 2-sided [-1.312 to -0.560] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Summary of Nicotine Equivalents Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of nicotine equivalents amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) for each metabolite were set to one-half of the LLOQ for the calculation of nicotine equivalents. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void). Nicotine equivalents (mg/g creatinine) = nicotine equivalents (μg/mL) x 100 / creatinine (mg/dL)
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | -1.783 (20.5643) | -25.070 (23.9100) | -13.053 (18.9294) | -67.749 (33.9247) | -45.240 (41.5952) | -95.808 (1.9997)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 0.870 (21.7462) | -22.036 (22.1901) | -11.641 (21.2360) | -68.537 (37.0327) | -51.521 (35.9795) | -96.968 (1.4462)

7. Secondary Outcome: Summary of 2-AN Amount Excreted and Absolute Change From Baseline (ng/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 2-aminonaphthalene (2-AN) amount excreted (ng/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (1.7 pg/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ng/24 hour
  Day -1 | 35.058 (14.7440) | 38.438 (16.5800) | 39.133 (20.5915) | 36.900 (18.4031) | 35.420 (13.9413) | 39.841 (17.9932)
  Day 5 | 33.753 (13.9940) | 21.422 (13.0808) | 21.325 (9.9158) | 2.760 (1.6132) | 2.085 (1.0846) | 2.410 (1.2299)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 35.786 (16.7327) | 20.031 (8.1023) | 20.709 (10.3490) | 2.757 (2.6274) | 1.777 (0.8171) | 2.849 (2.2411)
  Change from Baseline (Day 5) | -1.304 (8.4746) | -17.016 (15.3994) | -17.808 (19.0237) | -34.140 (18.8337) | -33.335 (13.4748) | -37.431 (18.0022)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | 0.728 (10.3513) | -18.505 (13.1224) | -18.424 (17.5363) | -33.896 (19.2124) | -33.997 (13.1827) | -36.606 (17.8281)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.470, 95% CI 2-sided [3.310 to 3.630] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.508, 95% CI 2-sided [3.348 to 3.668] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.891, 95% CI 2-sided [2.741 to 3.042] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.873, 95% CI 2-sided [2.719 to 3.027] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.928, 95% CI 2-sided [2.775 to 3.082] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.896, 95% CI 2-sided [2.742 to 3.049] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.864, 95% CI 2-sided [0.672 to 1.055] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.786, 95% CI 2-sided [0.592 to 0.981] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.641, 95% CI 2-sided [0.452 to 0.829] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.485, 95% CI 2-sided [0.290 to 0.680] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.747, 95% CI 2-sided [0.562 to 0.932] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.833, 95% CI 2-sided [0.645 to 1.021] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.579, 95% CI 2-sided [-0.889 to -0.268] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.635, 95% CI 2-sided [-0.949 to -0.321] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.542, 95% CI 2-sided [-0.853 to -0.231] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.613, 95% CI 2-sided [-0.924 to -0.301] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.606, 95% CI 2-sided [-2.959 to -2.253] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.722, 95% CI 2-sided [-3.078 to -2.366] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.829, 95% CI 2-sided [-3.177 to -2.481] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.024, 95% CI 2-sided [-3.378 to -2.669] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.144, 95% CI 2-sided [1.811 to 2.478] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.040, 95% CI 2-sided [1.701 to 2.379] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.181, 95% CI 2-sided [1.846 to 2.516] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.063, 95% CI 2-sided [1.725 to 2.400] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9705, Mixed Models Analysis; Mean Difference (Net) = 0.117, 95% CI 2-sided [-0.256 to 0.490] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -0.047, 95% CI 2-sided [-0.425 to 0.332] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9835, Mixed Models Analysis; Mean Difference (Net) = -0.106, 95% CI 2-sided [-0.475 to 0.263] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 2-AN amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.0854, Mixed Models Analysis; Mean Difference (Net) = -0.348, 95% CI 2-sided [-0.725 to 0.029] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Summary of 2-AN Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 2-aminonaphthalene (2-AN) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (1.7 pg/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | -0.214 (26.2880) | -41.725 (34.1635) | -29.316 (83.0987) | -90.186 (8.2459) | -93.792 (2.8305) | -93.291 (3.3952)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 4.815 (36.9328) | -44.657 (15.4429) | -39.152 (34.9209) | -90.671 (9.5679) | -94.813 (1.9651) | -92.289 (5.3199)

9. Secondary Outcome: Summary of 4-ABP Amount Excreted and Absolute Change From Baseline (ng/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 4-aminobiphenyl (4-ABP) amount excreted (ng/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (1.5 pg/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ng/24 hour
  Day -1 | 23.544 (7.4856) | 27.465 (11.1330) | 26.519 (9.2829) | 25.848 (11.3291) | 24.833 (8.8138) | 26.229 (7.3619)
  Day 5 | 21.449 (8.2875) | 15.684 (9.7048) | 16.673 (6.8533) | 3.785 (1.8918) | 3.692 (1.5741) | 3.826 (2.0856)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 21.700 (8.5794) | 14.315 (4.8816) | 15.567 (6.1982) | 3.484 (1.7674) | 3.422 (1.2121) | 3.577 (1.2299)
  Change from Baseline (Day 5) | -2.095 (5.7359) | -11.782 (10.5603) | -9.846 (7.3757) | -22.063 (11.0772) | -21.140 (7.9655) | -22.403 (7.0583)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -1.845 (6.5921) | -13.155 (7.7979) | -10.951 (7.0304) | -22.223 (11.3969) | -21.704 (8.2641) | -22.419 (7.2026)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.028, 95% CI 2-sided [2.901 to 3.154] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.034, 95% CI 2-sided [2.927 to 3.141] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.603, 95% CI 2-sided [2.483 to 2.722] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.567, 95% CI 2-sided [2.465 to 2.670] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.716, 95% CI 2-sided [2.595 to 2.838] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.643, 95% CI 2-sided [2.541 to 2.746] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.235, 95% CI 2-sided [1.083 to 1.386] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.174, 95% CI 2-sided [1.045 to 1.304] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.219, 95% CI 2-sided [1.070 to 1.368] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.176, 95% CI 2-sided [1.046 to 1.306] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.176, 95% CI 2-sided [1.029 to 1.322] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.174, 95% CI 2-sided [1.049 to 1.300] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.425, 95% CI 2-sided [-0.669 to -0.181] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.467, 95% CI 2-sided [-0.677 to -0.256] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0052, Mixed Models Analysis; Mean Difference (Net) = -0.311, 95% CI 2-sided [-0.556 to -0.066] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.391, 95% CI 2-sided [-0.600 to -0.182] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.793, 95% CI 2-sided [-2.070 to -1.516] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.859, 95% CI 2-sided [-2.098 to -1.621] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.809, 95% CI 2-sided [-2.082 to -1.535] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.858, 95% CI 2-sided [-2.096 to -1.621] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.427, 95% CI 2-sided [1.166 to 1.688] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.393, 95% CI 2-sided [1.166 to 1.620] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.541, 95% CI 2-sided [1.278 to 1.803] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.469, 95% CI 2-sided [1.243 to 1.695] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9987, Mixed Models Analysis; Mean Difference (Net) = 0.059, 95% CI 2-sided [-0.233 to 0.351] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.000, 95% CI 2-sided [-0.253 to 0.254] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9999, Mixed Models Analysis; Mean Difference (Net) = 0.043, 95% CI 2-sided [-0.246 to 0.332] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 4-ABP amount excreted (ng/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.002, 95% CI 2-sided [-0.251 to 0.254] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Summary of 4-ABP Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 4-aminobiphenyl (4-ABP) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (1.5 pg/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | -7.609 (26.3983) | -40.399 (31.8530) | -34.438 (20.0016) | -83.203 (9.1553) | -84.690 (6.4161) | -84.782 (8.1574)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -5.403 (40.5212) | -44.837 (13.1354) | -38.874 (19.1985) | -84.141 (9.2230) | -85.226 (5.6972) | -85.492 (6.0029)

11. Secondary Outcome: Summary of HEMA Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 2-hydroxyethyl mercapturic acid (HEMA) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.2 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 13.637 (6.7273) | 17.845 (12.7203) | 15.730 (12.9229) | 17.668 (15.0939) | 20.015 (12.5156) | 17.608 (12.9125)
  Day 5 | 11.473 (6.2511) | 12.822 (9.6015) | 10.819 (6.9893) | 8.768 (6.5494) | 11.119 (6.9600) | 8.115 (5.1282)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 11.316 (5.6391) | 12.475 (8.8931) | 10.571 (6.4028) | 8.393 (6.3959) | 10.289 (5.6391) | 9.284 (7.0913)
  Change from Baseline (Day 5) | -2.165 (4.4766) | -5.023 (6.7570) | -4.910 (7.9708) | -8.900 (12.5444) | -8.897 (9.5751) | -9.493 (9.9659)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -2.322 (4.9621) | -5.806 (7.8918) | -5.158 (8.3038) | -9.383 (12.2677) | -9.865 (10.8247) | -8.385 (10.4569)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.407, 95% CI 2-sided [2.283 to 2.531] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.398, 95% CI 2-sided [2.253 to 2.543] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.303, 95% CI 2-sided [2.187 to 2.420] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.250, 95% CI 2-sided [2.112 to 2.389] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.285, 95% CI 2-sided [2.166 to 2.404] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.272, 95% CI 2-sided [2.133 to 2.412] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.992, 95% CI 2-sided [1.844 to 2.140] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.894, 95% CI 2-sided [1.719 to 2.069] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.102, 95% CI 2-sided [1.955 to 2.248] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.075, 95% CI 2-sided [1.900 to 2.250] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.890, 95% CI 2-sided [1.746 to 2.033] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.944, 95% CI 2-sided [1.775 to 2.114] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.8674, Mixed Models Analysis; Mean Difference (Net) = -0.104, 95% CI 2-sided [-0.345 to 0.137] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.6519, Mixed Models Analysis; Mean Difference (Net) = -0.148, 95% CI 2-sided [-0.429 to 0.133] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.7301, Mixed Models Analysis; Mean Difference (Net) = -0.122, 95% CI 2-sided [-0.363 to 0.119] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.8076, Mixed Models Analysis; Mean Difference (Net) = -0.126, 95% CI 2-sided [-0.405 to 0.154] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0004, Mixed Models Analysis; Mean Difference (Net) = -0.415, 95% CI 2-sided [-0.689 to -0.142] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = -0.504, 95% CI 2-sided [-0.822 to -0.185] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0183, Mixed Models Analysis; Mean Difference (Net) = -0.306, 95% CI 2-sided [-0.578 to -0.034] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0443, Mixed Models Analysis; Mean Difference (Net) = -0.323, 95% CI 2-sided [-0.641 to -0.005] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = 0.414, 95% CI 2-sided [0.155 to 0.672] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.0454, Mixed Models Analysis; Mean Difference (Net) = 0.306, 95% CI 2-sided [0.004 to 0.608] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.0004, Mixed Models Analysis; Mean Difference (Net) = 0.396, 95% CI 2-sided [0.136 to 0.655] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.0261, Mixed Models Analysis; Mean Difference (Net) = 0.328, 95% CI 2-sided [0.026 to 0.630] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9455, Mixed Models Analysis; Mean Difference (Net) = 0.102, 95% CI 2-sided [-0.187 to 0.392] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.9999, Mixed Models Analysis; Mean Difference (Net) = -0.050, 95% CI 2-sided [-0.387 to 0.287] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.2633, Mixed Models Analysis; Mean Difference (Net) = 0.212, 95% CI 2-sided [-0.074 to 0.498] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: HEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.8769, Mixed Models Analysis; Mean Difference (Net) = 0.130, 95% CI 2-sided [-0.205 to 0.465] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Summary of HEMA Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 2-hydroxyethyl mercapturic acid (HEMA) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.2 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | -9.584 (33.1121) | -22.916 (29.9492) | -21.244 (28.9372) | -39.163 (28.8018) | -37.608 (30.2394) | -48.200 (21.7805)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -8.742 (37.0142) | -26.992 (30.6250) | -21.940 (27.9936) | -43.496 (27.6577) | -37.026 (42.9784) | -40.293 (31.7717)

13. Secondary Outcome: Summary of CEMA Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 2-cyanoethylmercapturic acid (CEMA) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.25 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 252.743 (95.7493) | 262.505 (105.5709) | 283.673 (126.9412) | 265.581 (136.7904) | 255.488 (89.9874) | 255.411 (88.5824)
  Day 5 | 235.071 (83.9199) | 156.653 (67.8784) | 169.389 (75.8871) | 36.060 (18.6284) | 37.816 (16.3173) | 36.648 (17.0519)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 242.647 (100.2513) | 162.257 (75.7299) | 169.996 (77.5677) | 34.356 (24.5937) | 33.700 (14.6351) | 35.135 (16.9140)
  Change from Baseline (Day 5) | -17.672 (59.2731) | -105.852 (61.4166) | -114.284 (90.2413) | -229.521 (123.5594) | -217.672 (78.9090) | -218.763 (82.4287)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -10.097 (61.2663) | -99.937 (66.7027) | -113.677 (83.6432) | -231.814 (130.7230) | -222.204 (82.1047) | -216.801 (79.5800)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.417, 95% CI 2-sided [5.315 to 5.520] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.436, 95% CI 2-sided [5.324 to 5.548] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.957, 95% CI 2-sided [4.860 to 5.053] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.974, 95% CI 2-sided [4.867 to 5.081] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.984, 95% CI 2-sided [4.886 to 5.082] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.975, 95% CI 2-sided [4.868 to 5.082] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.490, 95% CI 2-sided [3.367 to 3.612] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.347, 95% CI 2-sided [3.212 to 3.483] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.539, 95% CI 2-sided [3.418 to 3.660] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.419, 95% CI 2-sided [3.284 to 3.554] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.492, 95% CI 2-sided [3.373 to 3.611] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.437, 95% CI 2-sided [3.306 to 3.568] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.461, 95% CI 2-sided [-0.660 to -0.262] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.462, 95% CI 2-sided [-0.679 to -0.244] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.433, 95% CI 2-sided [-0.633 to -0.233] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.461, 95% CI 2-sided [-0.678 to -0.244] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.928, 95% CI 2-sided [-2.154 to -1.701] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.089, 95% CI 2-sided [-2.336 to -1.842] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.879, 95% CI 2-sided [-2.102 to -1.656] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.017, 95% CI 2-sided [-2.262 to -1.772] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.465, 95% CI 2-sided [1.250 to 1.679] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.537, 95% CI 2-sided [1.303 to 1.772] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.492, 95% CI 2-sided [1.277 to 1.707] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (PP Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.538, 95% CI 2-sided [1.304 to 1.772] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (PP Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -0.003, 95% CI 2-sided [-0.242 to 0.237] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (PP Population); p = 0.9399, Mixed Models Analysis; Mean Difference (Net) = -0.090, 95% CI 2-sided [-0.351 to 0.172] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (PP Population); p = 0.9993, Mixed Models Analysis; Mean Difference (Net) = 0.047, 95% CI 2-sided [-0.190 to 0.283] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (PP Population); Test type: Equivalence — Null hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: CEMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (PP Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -0.018, 95% CI 2-sided [-0.278 to 0.242] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Summary of CEMA Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 2-cyanoethylmercapturic acid (CEMA) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.25 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | -1.763 (32.1658) | -39.043 (15.6110) | -37.945 (16.1205) | -85.459 (5.5487) | -85.106 (4.6221) | -84.942 (6.4947)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -0.027 (35.0628) | -37.125 (15.0814) | -38.185 (15.7489) | -86.194 (10.0102) | -86.538 (3.8480) | -85.900 (5.1478)

15. Secondary Outcome: Summary of S-PMA Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of S-phenyl mercapturic acid (S-PMA) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.02 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 6.961 (3.8113) | 8.075 (5.6048) | 9.077 (5.8678) | 8.540 (5.0936) | 6.542 (3.7377) | 6.756 (5.0746)
  Day 5 | 6.935 (3.7971) | 4.792 (3.4372) | 5.559 (3.9536) | 0.557 (0.5157) | 0.377 (0.1812) | 0.511 (0.3146)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 6.808 (3.6133) | 4.820 (3.0674) | 5.358 (3.7852) | 0.482 (0.4835) | 0.319 (0.1300) | 0.458 (0.2561)
  Change from Baseline (Day 5) | -0.026 (1.8063) | -3.283 (2.7294) | -3.518 (4.0242) | -7.984 (4.9245) | -6.165 (3.6217) | -6.246 (4.8651)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -0.153 (2.0043) | -3.379 (3.1614) | -3.719 (3.6616) | -7.948 (5.0623) | -6.382 (3.6273) | -6.239 (4.9976)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.805, 95% CI 2-sided [1.639 to 1.971] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.788, 95% CI 2-sided [1.622 to 1.954] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.290, 95% CI 2-sided [1.145 to 1.462] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.304, 95% CI 2-sided [1.134 to 1.447] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.353, 95% CI 2-sided [1.194 to 1.513] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.313, 95% CI 2-sided [1.153 to 1.472] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.956, 95% CI 2-sided [-1.155 to -0.756] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.114, 95% CI 2-sided [-1.315 to -0.913] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.999, 95% CI 2-sided [-1.195 to -0.803] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.164, 95% CI 2-sided [-1.364 to -0.964] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.775, 95% CI 2-sided [-0.969 to -0.582] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.795, 95% CI 2-sided [-0.990 to -0.600] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = -0.514, 95% CI 2-sided [-0.836 to -0.193] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0005, Mixed Models Analysis; Mean Difference (Net) = -0.484, 95% CI 2-sided [-0.808 to -0.160] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0014, Mixed Models Analysis; Mean Difference (Net) = -0.452, 95% CI 2-sided [-0.775 to -0.128] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0007, Mixed Models Analysis; Mean Difference (Net) = -0.475, 95% CI 2-sided [-0.799 to -0.152] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.760, 95% CI 2-sided [-3.127 to -2.394] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.902, 95% CI 2-sided [-3.271 to -2.533] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.804, 95% CI 2-sided [-3.165 to -2.443] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.952, 95% CI 2-sided [-3.317 to -2.587] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.066, 95% CI 2-sided [1.719 to 2.413] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.099, 95% CI 2-sided [1.748 to 2.449] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.129, 95% CI 2-sided [1.779 to 2.478] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.107, 95% CI 2-sided [1.756 to 2.459] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.7678, Mixed Models Analysis; Mean Difference (Net) = -0.180, 95% CI 2-sided [-0.569 to 0.209] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.1691, Mixed Models Analysis; Mean Difference (Net) = -0.319, 95% CI 2-sided [-0.711 to 0.073] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.5178, Mixed Models Analysis; Mean Difference (Net) = -0.224, 95% CI 2-sided [-0.606 to 0.158] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: S-PMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.0699, Mixed Models Analysis; Mean Difference (Net) = -0.369, 95% CI 2-sided [-0.757 to 0.018] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Summary of S-PMA Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of S-phenyl mercapturic acid (S-PMA) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.02 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | 0.414 (27.7146) | -39.223 (16.7927) | -32.680 (44.7678) | -92.361 (5.6169) | -92.666 (5.5760) | -89.785 (7.9606)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -0.440 (27.6623) | -37.688 (15.2518) | -36.710 (33.5234) | -92.651 (7.7763) | -93.659 (5.2551) | -90.037 (8.0553)

17. Secondary Outcome: Summary of 3-HMPMA Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 3-hydroxy-1-methylpropylmercapturic acid (3-HMPMA) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (5 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 550.337 (205.3039) | 566.207 (212.2527) | 620.251 (282.7648) | 606.423 (388.1189) | 569.736 (236.5974) | 563.298 (237.6972)
  Day 5 | 508.316 (206.5741) | 354.525 (133.4293) | 404.976 (183.1641) | 167.136 (103.8973) | 144.751 (65.9291) | 141.885 (80.2953)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 521.141 (217.2385) | 368.736 (160.2715) | 383.715 (158.6928) | 150.400 (63.8041) | 157.595 (79.8494) | 155.132 (75.3979)
  Change from Baseline (Day 5) | -42.021 (124.9105) | -211.682 (131.0495) | -215.275 (189.0406) | -439.287 (355.2849) | -424.984 (215.2851) | -421.414 (213.6181)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -29.196 (131.9289) | -193.629 (132.1995) | -236.535 (185.1107) | -455.759 (392.8206) | -414.706 (229.5738) | -411.417 (194.8371)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 6.177, 95% CI 2-sided [6.062 to 6.292] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 6.197, 95% CI 2-sided [6.082 to 6.312] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.798, 95% CI 2-sided [5.690 to 5.906] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.820, 95% CI 2-sided [5.710 to 5.930] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.863, 95% CI 2-sided [5.753 to 5.974] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.816, 95% CI 2-sided [5.706 to 5.927] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.947, 95% CI 2-sided [4.809 to 5.084] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.913, 95% CI 2-sided [4.774 to 5.052] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.862, 95% CI 2-sided [4.727 to 4.998] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.938, 95% CI 2-sided [4.799 to 5.076] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.826, 95% CI 2-sided [4.693 to 4.959] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.902, 95% CI 2-sided [4.767 to 5.037] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.379, 95% CI 2-sided [-0.602 to -0.156] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.376, 95% CI 2-sided [-0.601 to -0.152] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0014, Mixed Models Analysis; Mean Difference (Net) = -0.314, 95% CI 2-sided [-0.537 to -0.090] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.381, 95% CI 2-sided [-0.604 to -0.157] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.230, 95% CI 2-sided [-1.484 to -0.977] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.284, 95% CI 2-sided [-1.539 to -1.029] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.315, 95% CI 2-sided [-1.564 to -1.065] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.259, 95% CI 2-sided [-1.512 to -1.006] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.972, 95% CI 2-sided [0.732 to 1.211] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.918, 95% CI 2-sided [0.676 to 1.161] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.037, 95% CI 2-sided [0.797 to 1.278] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.914, 95% CI 2-sided [0.672 to 1.156] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.7939, Mixed Models Analysis; Mean Difference (Net) = 0.121, 95% CI 2-sided [-0.147 to 0.388] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.011, 95% CI 2-sided [-0.260 to 0.281] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.036, 95% CI 2-sided [-0.228 to 0.301] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HMPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.036, 95% CI 2-sided [-0.233 to 0.305] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Summary of 3-HMPMA Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 3-hydroxy-1-methylpropylmercapturic acid (3-HMPMA) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (5 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | -5.743 (22.6960) | -35.546 (13.9889) | -32.157 (17.5366) | -68.831 (18.5627) | -72.980 (12.2613) | -73.991 (12.7785)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -3.562 (25.6505) | -33.002 (17.2920) | -35.002 (15.4967) | -68.732 (19.6288) | -70.424 (15.9381) | -72.466 (9.0818)

19. Secondary Outcome: Summary of 3-HPMA Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 3-hydroxypropylmercapturic acid (3-HPMA) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (25 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 1743.226 (668.1382) | 1766.765 (615.6747) | 1986.391 (853.8727) | 1865.738 (901.8706) | 1811.893 (878.2589) | 1922.765 (697.3324)
  Day 5 | 1677.258 (665.1729) | 1043.324 (409.5555) | 1201.051 (542.2406) | 433.971 (295.7202) | 460.103 (391.5957) | 471.823 (210.0711)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 1658.754 (609.9999) | 1047.861 (369.5717) | 1152.712 (512.4255) | 384.725 (186.4687) | 414.764 (193.2655) | 465.606 (181.1420)
  Change from Baseline (Day 5) | -65.969 (393.3398) | -723.442 (409.5358) | -785.340 (505.9671) | -1431.767 (841.9879) | -1351.790 (761.5792) | -1450.942 (571.8160)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -84.472 (405.0119) | -715.263 (368.4390) | -833.680 (621.2865) | -1485.874 (894.8234) | -1442.549 (862.2948) | -1455.899 (646.1344)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 7.367, 95% CI 2-sided [7.250 to 7.485] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 7.368, 95% CI 2-sided [7.251 to 7.485] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 6.883, 95% CI 2-sided [6.773 to 6.994] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 6.892, 95% CI 2-sided [6.780 to 7.004] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 6.942, 95% CI 2-sided [6.829 to 7.054] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 6.896, 95% CI 2-sided [6.784 to 7.008] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.879, 95% CI 2-sided [5.739 to 6.019] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.804, 95% CI 2-sided [5.662 to 5.946] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.916, 95% CI 2-sided [5.778 to 6.054] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.917, 95% CI 2-sided [5.775 to 6.058] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 6.017, 95% CI 2-sided [5.881 to 6.153] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 6.012, 95% CI 2-sided [5.874 to 6.149] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.484, 95% CI 2-sided [-0.711 to -0.257] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.476, 95% CI 2-sided [-0.705 to -0.248] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.426, 95% CI 2-sided [-0.654 to -0.198] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.472, 95% CI 2-sided [-0.701 to -0.244] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.489, 95% CI 2-sided [-1.747 to -1.230] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.564, 95% CI 2-sided [-1.825 to -1.304] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.451, 95% CI 2-sided [-1.706 to -1.197] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.452, 95% CI 2-sided [-1.710 to -1.193] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.866, 95% CI 2-sided [0.622 to 1.110] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.880, 95% CI 2-sided [0.633 to 1.128] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.924, 95% CI 2-sided [0.680 to 1.169] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.884, 95% CI 2-sided [0.638 to 1.131] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.6800, Mixed Models Analysis; Mean Difference (Net) = -0.138, 95% CI 2-sided [-0.411 to 0.134] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.2371, Mixed Models Analysis; Mean Difference (Net) = -0.208, 95% CI 2-sided [-0.483 to 0.068] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9133, Mixed Models Analysis; Mean Difference (Net) = -0.101, 95% CI 2-sided [-0.371 to 0.169] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 3-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.9432, Mixed Models Analysis; Mean Difference (Net) = -0.095, 95% CI 2-sided [-0.370 to 0.180] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Summary of 3-HPMA Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 3-hydroxypropylmercapturic acid (3-HPMA) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (25 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | -1.420 (24.6382) | -39.382 (16.8251) | -37.881 (14.6021) | -75.303 (13.2868) | -74.412 (14.4248) | -74.897 (7.6082)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -1.110 (25.6542) | -39.328 (10.6349) | -39.461 (16.1768) | -76.922 (13.0070) | -74.522 (13.5851) | -74.238 (9.0407)

21. Secondary Outcome: Summary of 2-HPMA Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 2-hydroxypropyl-mercapturic acid (2-HPMA) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (2.5 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 105.297 (54.5963) | 110.378 (62.4698) | 113.258 (64.2108) | 116.041 (64.3856) | 108.420 (63.0178) | 115.231 (54.4428)
  Day 5 | 106.168 (59.9458) | 73.687 (45.6677) | 73.431 (32.8976) | 21.284 (7.7785) | 36.173 (40.3089) | 23.226 (7.9556)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 100.714 (51.4490) | 72.440 (39.9138) | 70.583 (31.1338) | 22.004 (9.4428) | 33.002 (18.4874) | 26.843 (9.3874)
  Change from Baseline (Day 5) | 0.871 (34.9551) | -36.691 (33.3048) | -39.827 (47.7576) | -94.758 (63.0836) | -72.247 (71.8521) | -92.006 (53.5034)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -4.583 (21.8338) | -39.574 (33.6340) | -42.675 (52.2138) | -93.636 (65.3517) | -77.317 (65.6904) | -89.342 (53.0876)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.513, 95% CI 2-sided [4.383 to 4.643] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.491, 95% CI 2-sided [4.371 to 4.610] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.150, 95% CI 2-sided [4.027 to 4.272] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.128, 95% CI 2-sided [4.014 to 4.242] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.176, 95% CI 2-sided [4.051 to 4.301] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.139, 95% CI 2-sided [4.024 to 4.254] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.997, 95% CI 2-sided [2.842 to 3.153] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.994, 95% CI 2-sided [2.849 to 3.138] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.317, 95% CI 2-sided [3.164 to 3.470] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.342, 95% CI 2-sided [3.199 to 3.486] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.036, 95% CI 2-sided [2.886 to 3.187] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.159, 95% CI 2-sided [3.019 to 3.299] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0008, Mixed Models Analysis; Mean Difference (Net) = -0.363, 95% CI 2-sided [-0.613 to -0.113] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = -0.362, 95% CI 2-sided [-0.595 to -0.129] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0026, Mixed Models Analysis; Mean Difference (Net) = -0.337, 95% CI 2-sided [-0.588 to -0.085] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0004, Mixed Models Analysis; Mean Difference (Net) = -0.351, 95% CI 2-sided [-0.584 to -0.118] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.515, 95% CI 2-sided [-1.800 to -1.230] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.497, 95% CI 2-sided [-1.762 to -1.231] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.196, 95% CI 2-sided [-1.477 to -0.915] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.148, 95% CI 2-sided [-1.410 to -0.886] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.113, 95% CI 2-sided [0.844 to 1.382] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.969, 95% CI 2-sided [0.717 to 1.221] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.139, 95% CI 2-sided [0.869 to 1.410] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.980, 95% CI 2-sided [0.728 to 1.231] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -0.039, 95% CI 2-sided [-0.340 to 0.262] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.5184, Mixed Models Analysis; Mean Difference (Net) = -0.166, 95% CI 2-sided [-0.447 to 0.115] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.0743, Mixed Models Analysis; Mean Difference (Net) = 0.280, 95% CI 2-sided [-0.017 to 0.578] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 2-HPMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.3889, Mixed Models Analysis; Mean Difference (Net) = 0.183, 95% CI 2-sided [-0.095 to 0.462] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Summary of 2-HPMA Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 2-hydroxypropyl-mercapturic acid (2-HPMA) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (2.5 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | 2.576 (35.0793) | -30.260 (22.7811) | -28.992 (20.1727) | -73.489 (21.9780) | -59.835 (42.1367) | -75.225 (16.1842)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -1.857 (20.6712) | -32.286 (15.7228) | -30.611 (19.9059) | -72.078 (24.0289) | -61.684 (33.6407) | -71.565 (20.1576)

23. Secondary Outcome: Summary of AAMA Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of N-acetyl-S-(2-carbamoylethyl)-l-cysteine (AAMA) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (10 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 205.752 (69.9796) | 213.840 (84.3383) | 234.379 (110.9685) | 179.355 (60.6867) | 203.156 (69.9106) | 212.299 (72.6566)
  Day 5 | 209.546 (92.1646) | 170.626 (87.7149) | 194.963 (78.8241) | 99.589 (70.9683) | 91.040 (46.5105) | 103.427 (61.1171)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 196.301 (78.9983) | 162.085 (77.9669) | 185.991 (85.8673) | 85.598 (53.8351) | 84.941 (36.0825) | 112.082 (48.2731)
  Change from Baseline (Day 5) | 3.794 (61.0286) | -43.214 (47.8198) | -39.416 (74.9528) | -79.766 (73.7312) | -112.116 (61.2701) | -108.872 (60.5423)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -9.451 (47.6276) | -53.542 (45.4159) | -48.387 (69.3531) | -96.049 (49.6356) | -122.821 (56.8629) | -96.887 (57.5065)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.264, 95% CI 2-sided [5.155 to 5.373] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.204, 95% CI 2-sided [5.106 to 5.302] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.005, 95% CI 2-sided [4.902 to 5.108] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.958, 95% CI 2-sided [4.864 to 5.051] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.114, 95% CI 2-sided [5.009 to 5.219] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.052, 95% CI 2-sided [4.958 to 5.146] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.539, 95% CI 2-sided [4.407 to 4.671] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.415, 95% CI 2-sided [4.295 to 4.534] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.431, 95% CI 2-sided [4.302 to 4.560] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.361, 95% CI 2-sided [4.243 to 4.480] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.486, 95% CI 2-sided [4.359 to 4.612] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 4.588, 95% CI 2-sided [4.473 to 4.703] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0073, Mixed Models Analysis; Mean Difference (Net) = -0.259, 95% CI 2-sided [-0.469 to -0.049] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0041, Mixed Models Analysis; Mean Difference (Net) = -0.246, 95% CI 2-sided [-0.438 to -0.055] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.3080, Mixed Models Analysis; Mean Difference (Net) = -0.150, 95% CI 2-sided [-0.361 to 0.061] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.1982, Mixed Models Analysis; Mean Difference (Net) = -0.152, 95% CI 2-sided [-0.343 to 0.039] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.725, 95% CI 2-sided [-0.965 to -0.486] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.790, 95% CI 2-sided [-1.008 to -0.571] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.833, 95% CI 2-sided [-1.069 to -0.597] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.843, 95% CI 2-sided [-1.059 to -0.627] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.520, 95% CI 2-sided [0.294 to 0.745] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.370, 95% CI 2-sided [0.163 to 0.577] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.628, 95% CI 2-sided [0.402 to 0.855] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.464, 95% CI 2-sided [0.257 to 0.670] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9984, Mixed Models Analysis; Mean Difference (Net) = 0.053, 95% CI 2-sided [-0.200 to 0.306] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.2491, Mixed Models Analysis; Mean Difference (Net) = -0.173, 95% CI 2-sided [-0.405 to 0.058] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9977, Mixed Models Analysis; Mean Difference (Net) = -0.054, 95% CI 2-sided [-0.304 to 0.195] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: AAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.0554, Mixed Models Analysis; Mean Difference (Net) = -0.227, 95% CI 2-sided [-0.456 to 0.003] — [estimate comment as in outcome 1, analysis 1]

24. Secondary Outcome: Summary of AAMA Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of N-acetyl-S-(2-carbamoylethyl)-l-cysteine (AAMA) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original Values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (10 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | 2.922 (27.1486) | -20.973 (22.5861) | -11.986 (25.3885) | -43.579 (35.6609) | -53.493 (21.2336) | -51.247 (20.0931)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -3.571 (22.7243) | -25.039 (17.9283) | -17.088 (22.3929) | -53.682 (18.2362) | -57.436 (15.7971) | -45.335 (20.0234)

25. Secondary Outcome: Summary of GAMA Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of N-acetyl-S-(2-carbamoyl-2-hydroxyethyl)-l-cysteine (GAMA) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (1 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 28.151 (7.9362) | 30.337 (9.1426) | 30.415 (12.2998) | 25.403 (7.9934) | 26.270 (9.0014) | 30.737 (10.1313)
  Day 5 | 28.123 (9.0482) | 24.988 (8.6134) | 26.343 (9.3111) | 15.898 (6.4032) | 15.080 (5.3359) | 17.982 (8.1223)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 27.310 (8.8508) | 24.808 (9.1001) | 25.701 (9.1838) | 14.184 (6.1136) | 14.272 (5.0565) | 18.856 (6.6119)
  Change from Baseline (Day 5) | -0.029 (6.6123) | -5.349 (6.0495) | -4.072 (8.5389) | -9.504 (8.2824) | -11.190 (7.8064) | -12.754 (7.9808)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -0.842 (5.6395) | -5.562 (5.0722) | -4.714 (8.9415) | -11.525 (7.7630) | -12.681 (7.5912) | -11.638 (7.8765)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.294, 95% CI 2-sided [3.208 to 3.379] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.262, 95% CI 2-sided [3.176 to 3.348] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.120, 95% CI 2-sided [3.039 to 3.202] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.099, 95% CI 2-sided [3.017 to 3.181] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.182, 95% CI 2-sided [3.100 to 3.264] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.149, 95% CI 2-sided [3.066 to 3.231] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.777, 95% CI 2-sided [2.673 to 2.881] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.651, 95% CI 2-sided [2.546 to 2.756] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.720, 95% CI 2-sided [2.618 to 2.823] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.649, 95% CI 2-sided [2.544 to 2.753] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.751, 95% CI 2-sided [2.651 to 2.851] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.819, 95% CI 2-sided [2.718 to 2.919] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0377, Mixed Models Analysis; Mean Difference (Net) = -0.173, 95% CI 2-sided [-0.340 to -0.006] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0643, Mixed Models Analysis; Mean Difference (Net) = -0.163, 95% CI 2-sided [-0.331 to 0.006] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.3875, Mixed Models Analysis; Mean Difference (Net) = -0.112, 95% CI 2-sided [-0.279 to 0.056] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.3725, Mixed Models Analysis; Mean Difference (Net) = -0.113, 95% CI 2-sided [-0.280 to 0.054] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.516, 95% CI 2-sided [-0.706 to -0.327] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.611, 95% CI 2-sided [-0.802 to -0.420] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.573, 95% CI 2-sided [-0.760 to -0.386] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.613, 95% CI 2-sided [-0.803 to -0.423] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.369, 95% CI 2-sided [0.190 to 0.548] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = 0.280, 95% CI 2-sided [0.099 to 0.462] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.431, 95% CI 2-sided [0.251 to 0.611] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.330, 95% CI 2-sided [0.149 to 0.511] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.026, 95% CI 2-sided [-0.176 to 0.228] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.1589, Mixed Models Analysis; Mean Difference (Net) = -0.168, 95% CI 2-sided [-0.371 to 0.036] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9999, Mixed Models Analysis; Mean Difference (Net) = -0.031, 95% CI 2-sided [-0.230 to 0.168] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: GAMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.1453, Mixed Models Analysis; Mean Difference (Net) = -0.170, 95% CI 2-sided [-0.372 to 0.032] — [estimate comment as in outcome 1, analysis 1]

26. Secondary Outcome: Summary of GAMA Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of N-acetyl-S-(2-carbamoyl-2-hydroxyethyl)-l-cysteine (GAMA) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (1 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | 2.015 (23.0063) | -16.449 (19.0682) | -9.361 (23.0900) | -34.427 (25.2883) | -39.251 (22.4238) | -40.803 (18.2548)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -1.515 (21.1321) | -18.456 (16.3993) | -11.236 (24.0586) | -43.200 (19.3353) | -44.682 (19.3080) | -36.587 (16.0285)

27. Secondary Outcome: Summary of 2-MHBMA Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 2-hydroxybutenyl-mercapturic acid (2-MHBMA) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.129 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 5.230 (4.3362) | 6.226 (6.0371) | 7.136 (6.3804) | 5.866 (4.1432) | 4.146 (3.8962) | 5.136 (4.5388)
  Day 5 | 5.126 (3.6876) | 3.287 (3.0863) | 3.703 (3.5055) | 0.142 (0.0714) | 0.186 (0.1141) | 0.259 (0.2148)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 5.284 (4.4769) | 3.406 (3.1052) | 4.128 (3.4363) | 0.183 (0.1539) | 0.188 (0.1097) | 0.216 (0.1532)
  Change from Baseline (Day 5) | -0.104 (1.9552) | -2.939 (3.4047) | -3.433 (4.1785) | -5.724 (4.1297) | -3.960 (3.8836) | -4.877 (4.5654)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | 0.054 (2.3432) | -2.995 (3.6985) | -3.008 (4.1064) | -5.913 (4.0535) | -4.102 (3.9316) | -4.971 (4.6010)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.085, 95% CI 2-sided [0.788 to 1.382] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.104, 95% CI 2-sided [0.807 to 1.400] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.606, 95% CI 2-sided [0.326 to 0.886] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p = 0.0011, Mixed Models Analysis; Mean Difference (Net) = 0.476, 95% CI 2-sided [0.192 to 0.760] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p = 0.0006, Mixed Models Analysis; Mean Difference (Net) = 0.505, 95% CI 2-sided [0.219 to 0.790] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.775, 95% CI 2-sided [0.490 to 1.060] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.116, 95% CI 2-sided [-2.472 to -1.761] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.016, 95% CI 2-sided [-2.376 to -1.656] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.605, 95% CI 2-sided [-1.958 to -1.253] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.642, 95% CI 2-sided [-2.003 to -1.282] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.578, 95% CI 2-sided [-1.922 to -1.234] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.726, 95% CI 2-sided [-2.074 to -1.378] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.1579, Mixed Models Analysis; Mean Difference (Net) = -0.479, 95% CI 2-sided [-1.054 to 0.097] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0260, Mixed Models Analysis; Mean Difference (Net) = -0.628, 95% CI 2-sided [-1.207 to -0.048] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0483, Mixed Models Analysis; Mean Difference (Net) = -0.580, 95% CI 2-sided [-1.158 to -0.003] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.5842, Mixed Models Analysis; Mean Difference (Net) = -0.329, 95% CI 2-sided [-0.906 to 0.249] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.201, 95% CI 2-sided [-3.856 to -2.546] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.119, 95% CI 2-sided [-3.779 to -2.460] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.690, 95% CI 2-sided [-3.338 to -2.043] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.746, 95% CI 2-sided [-3.402 to -2.090] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.184, 95% CI 2-sided [1.565 to 2.803] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.202, 95% CI 2-sided [1.576 to 2.828] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.083, 95% CI 2-sided [1.461 to 2.704] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.501, 95% CI 2-sided [1.876 to 3.126] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.2085, Mixed Models Analysis; Mean Difference (Net) = -0.538, 95% CI 2-sided [-1.231 to 0.154] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.8557, Mixed Models Analysis; Mean Difference (Net) = -0.289, 95% CI 2-sided [-0.988 to 0.410] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -0.027, 95% CI 2-sided [-0.713 to 0.658] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 2-MHBMA amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.084, 95% CI 2-sided [-0.612 to 0.780] — [estimate comment as in outcome 1, analysis 1]

28. Secondary Outcome: Summary of 2-MHBMA Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 2-hydroxybutenyl-mercapturic acid (2-MHBMA) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.129 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | 89.466 (362.5275) | 39.458 (291.2398) | -3.704 (164.5239) | -82.576 (35.6633) | -66.761 (48.4733) | -50.591 (124.5982)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 97.272 (337.2550) | 28.617 (287.5681) | 66.188 (460.0304) | -76.231 (76.9824) | -68.019 (49.9841) | -72.699 (48.5745)

29. Secondary Outcome: Summary of 2-OHFLe Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 2-OH-Fluorene (2-OHFLe) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.1 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 27
ug/24 hour
  Day -1 | 6.013 (5.5242) | 6.453 (4.1583) | 4.947 (4.2710) | 5.424 (4.1109) | 8.101 (16.9678) | 4.852 (2.3571)
  Day 5: number analyzed (Participants) | 38 | 42 | 40 | 26 | 27 | 27
  Day 5 | 5.535 (5.5502) | 6.002 (14.2979) | 5.006 (10.0199) | 2.857 (2.6235) | 2.879 (4.0524) | 2.101 (1.2935)
  Day 7: number analyzed (Participants) | 37 | 40 | 41 | 25 | 25 | 26
  Day 7 | 5.471 (4.9675) | 4.029 (4.2137) | 3.219 (3.6982) | 2.238 (2.5664) | 2.493 (3.5417) | 2.046 (2.1506)
  Change from Baseline (Day 5): number analyzed (Participants) | 38 | 42 | 40 | 26 | 27 | 27
  Change from Baseline (Day 5) | -0.478 (5.8039) | -0.452 (15.4210) | -0.023 (9.1944) | -2.567 (4.2155) | -5.222 (16.0117) | -2.752 (2.0610)
  Change from Baseline (Day 7): number analyzed (Participants) | 37 | 40 | 41 | 25 | 25 | 26
  Change from Baseline (Day 7) | -0.668 (5.3174) | -2.386 (4.3279) | -1.728 (3.6338) | -3.176 (4.9330) | -5.989 (15.2327) | -2.710 (2.7968)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.081, 95% CI 2-sided [0.679 to 1.484] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.309, 95% CI 2-sided [0.902 to 1.716] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.996, 95% CI 2-sided [0.615 to 1.377] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = 0.728, 95% CI 2-sided [0.339 to 1.116] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.987, 95% CI 2-sided [0.593 to 1.381] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.865, 95% CI 2-sided [0.475 to 1.254] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p = 0.0768, Mixed Models Analysis; Mean Difference (Net) = 0.436, 95% CI 2-sided [-0.047 to 0.920] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p = 0.7155, Mixed Models Analysis; Mean Difference (Net) = 0.091, 95% CI 2-sided [-0.400 to 0.583] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p = 0.3282, Mixed Models Analysis; Mean Difference (Net) = 0.237, 95% CI 2-sided [-0.239 to 0.713] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p = 0.3578, Mixed Models Analysis; Mean Difference (Net) = -0.230, 95% CI 2-sided [-0.722 to 0.262] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p = 0.1638, Mixed Models Analysis; Mean Difference (Net) = 0.338, 95% CI 2-sided [-0.138 to 0.814] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p = 0.8384, Mixed Models Analysis; Mean Difference (Net) = -0.050, 95% CI 2-sided [-0.533 to 0.433] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -0.086, 95% CI 2-sided [-0.869 to 0.698] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.2808, Mixed Models Analysis; Mean Difference (Net) = -0.581, 95% CI 2-sided [-1.377 to 0.214] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -0.095, 95% CI 2-sided [-0.887 to 0.698] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.6018, Mixed Models Analysis; Mean Difference (Net) = -0.444, 95% CI 2-sided [-1.237 to 0.349] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.2935, Mixed Models Analysis; Mean Difference (Net) = -0.645, 95% CI 2-sided [-1.536 to 0.246] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0023, Mixed Models Analysis; Mean Difference (Net) = -1.218, 95% CI 2-sided [-2.120 to -0.315] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0669, Mixed Models Analysis; Mean Difference (Net) = -0.844, 95% CI 2-sided [-1.723 to 0.035] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.539, 95% CI 2-sided [-2.438 to -0.640] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.2120, Mixed Models Analysis; Mean Difference (Net) = 0.658, 95% CI 2-sided [-0.192 to 1.509] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.0993, Mixed Models Analysis; Mean Difference (Net) = 0.778, 95% CI 2-sided [-0.087 to 1.642] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.2347, Mixed Models Analysis; Mean Difference (Net) = 0.649, 95% CI 2-sided [-0.211 to 1.509] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.0320, Mixed Models Analysis; Mean Difference (Net) = 0.915, 95% CI 2-sided [0.052 to 1.778] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.099, 95% CI 2-sided [-0.849 to 1.047] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.9999, Mixed Models Analysis; Mean Difference (Net) = 0.141, 95% CI 2-sided [-0.820 to 1.103] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -0.101, 95% CI 2-sided [-1.038 to 0.837] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 2-OHFLe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.9995, Mixed Models Analysis; Mean Difference (Net) = -0.180, 95% CI 2-sided [-1.139 to 0.779] — [estimate comment as in outcome 1, analysis 1]

30. Secondary Outcome: Summary of 2-OHFLe Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 2-OH-Fluorene (2-OHFLe) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.1 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 27
percentage of change
  Day 5: number analyzed (Participants) | 38 | 42 | 40 | 26 | 27 | 27
  Day 5 | 12.958 (105.7554) | 5043.768 (32905.9569) | 178.037 (1045.5731) | -45.034 (38.3930) | -37.094 (118.0482) | -52.455 (32.2698)
  Day 7: number analyzed (Participants) | 37 | 40 | 41 | 25 | 25 | 26
  Day 7 | 15.496 (81.6064) | 503.991 (3454.7322) | 272.425 (1374.3325) | -48.971 (54.0298) | -63.094 (41.9257) | -54.026 (57.9650)

31. Secondary Outcome: Summary of 2-Naphthol Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 2-Naphthol amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.10 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 26.351 (13.4453) | 28.168 (9.0786) | 28.246 (12.6762) | 27.688 (12.7029) | 26.292 (8.6468) | 24.827 (9.7689)
  Day 5 | 23.047 (9.2844) | 16.141 (7.9059) | 16.385 (5.7688) | 6.559 (3.8649) | 6.407 (5.0282) | 7.299 (8.1699)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 23.191 (8.1002) | 16.228 (8.2504) | 15.475 (7.1820) | 6.670 (4.5266) | 5.436 (4.3673) | 8.216 (8.9779)
  Change from Baseline (Day 5) | -3.304 (13.7567) | -12.027 (6.3192) | -11.860 (11.0884) | -21.129 (12.6944) | -19.885 (8.2403) | -17.527 (8.9468)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -3.160 (13.3625) | -11.651 (5.1880) | -12.771 (10.2647) | -20.747 (13.6498) | -20.326 (9.2076) | -16.367 (8.8314)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.120, 95% CI 2-sided [2.964 to 3.276] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.141, 95% CI 2-sided [2.953 to 3.328] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.658, 95% CI 2-sided [2.511 to 2.806] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.638, 95% CI 2-sided [2.458 to 2.817] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.754, 95% CI 2-sided [2.604 to 2.903] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 2.652, 95% CI 2-sided [2.471 to 2.832] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.703, 95% CI 2-sided [1.517 to 1.889] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.637, 95% CI 2-sided [1.410 to 1.865] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.656, 95% CI 2-sided [1.472 to 1.839] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.485, 95% CI 2-sided [1.259 to 1.711] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.713, 95% CI 2-sided [1.532 to 1.895] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.617, 95% CI 2-sided [1.397 to 1.837] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = -0.462, 95% CI 2-sided [-0.766 to -0.158] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0018, Mixed Models Analysis; Mean Difference (Net) = -0.503, 95% CI 2-sided [-0.867 to -0.139] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0089, Mixed Models Analysis; Mean Difference (Net) = -0.366, 95% CI 2-sided [-0.670 to -0.062] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0025, Mixed Models Analysis; Mean Difference (Net) = -0.489, 95% CI 2-sided [-0.851 to -0.126] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.417, 95% CI 2-sided [-1.762 to -1.072] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.504, 95% CI 2-sided [-1.916 to -1.091] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.464, 95% CI 2-sided [-1.804 to -1.125] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.656, 95% CI 2-sided [-2.065 to -1.247] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.945, 95% CI 2-sided [0.617 to 1.273] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.021, 95% CI 2-sided [0.628 to 1.413] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.041, 95% CI 2-sided [0.712 to 1.369] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.035, 95% CI 2-sided [0.644 to 1.426] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -0.010, 95% CI 2-sided [-0.376 to 0.355] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.020, 95% CI 2-sided [-0.417 to 0.457] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9999, Mixed Models Analysis; Mean Difference (Net) = -0.058, 95% CI 2-sided [-0.418 to 0.303] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 2-Naphthol amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.9669, Mixed Models Analysis; Mean Difference (Net) = -0.132, 95% CI 2-sided [-0.566 to 0.301] — [estimate comment as in outcome 1, analysis 1]

32. Secondary Outcome: Summary of 2-Naphthol Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 2-Naphthol amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.10 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | -2.871 (48.4874) | -42.250 (17.7416) | -35.217 (25.6833) | -72.375 (20.2036) | -74.880 (16.3832) | -72.152 (20.3724)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -3.848 (33.7807) | -42.498 (16.2147) | -40.149 (24.8026) | -70.911 (23.8688) | -77.080 (18.5790) | -69.892 (26.9968)

33. Secondary Outcome: Summary of 1-OHPhe Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 1-OH-Phenanthrene (1-OHPhe) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.005 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 0.291 (0.1655) | 0.325 (0.1332) | 0.324 (0.1591) | 0.342 (0.1495) | 0.273 (0.1560) | 0.348 (0.1870)
  Day 5 | 0.278 (0.1902) | 0.206 (0.1019) | 0.214 (0.0966) | 0.147 (0.1357) | 0.101 (0.0567) | 0.131 (0.0617)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 0.273 (0.1779) | 0.190 (0.0833) | 0.190 (0.1011) | 0.126 (0.0827) | 0.095 (0.0546) | 0.149 (0.0923)
  Change from Baseline (Day 5) | -0.013 (0.1110) | -0.119 (0.1104) | -0.110 (0.1535) | -0.195 (0.2001) | -0.172 (0.1313) | -0.217 (0.1672)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -0.018 (0.1123) | -0.133 (0.0954) | -0.134 (0.1253) | -0.209 (0.1597) | -0.182 (0.1308) | -0.185 (0.1665)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.442, 95% CI 2-sided [-1.604 to -1.279] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.413, 95% CI 2-sided [-1.576 to -1.251] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.754, 95% CI 2-sided [-1.907 to -1.600] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.816, 95% CI 2-sided [-1.972 to -1.659] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.654, 95% CI 2-sided [-1.810 to -1.498] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.829, 95% CI 2-sided [-1.986 to -1.673] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.184, 95% CI 2-sided [-2.379 to -1.989] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.270, 95% CI 2-sided [-2.468 to -2.071] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.413, 95% CI 2-sided [-2.607 to -2.219] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.349, 95% CI 2-sided [-2.549 to -2.149] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.227, 95% CI 2-sided [-2.416 to -2.038] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.154, 95% CI 2-sided [-2.345 to -1.962] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0552, Mixed Models Analysis; Mean Difference (Net) = -0.312, 95% CI 2-sided [-0.628 to 0.004] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0055, Mixed Models Analysis; Mean Difference (Net) = -0.402, 95% CI 2-sided [-0.722 to -0.083] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.3834, Mixed Models Analysis; Mean Difference (Net) = -0.212, 95% CI 2-sided [-0.530 to 0.105] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0033, Mixed Models Analysis; Mean Difference (Net) = -0.416, 95% CI 2-sided [-0.734 to -0.099] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.743, 95% CI 2-sided [-1.103 to -0.382] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.857, 95% CI 2-sided [-1.220 to -0.493] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.971, 95% CI 2-sided [-1.327 to -0.616] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.936, 95% CI 2-sided [-1.298 to -0.574] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.0016, Mixed Models Analysis; Mean Difference (Net) = 0.473, 95% CI 2-sided [0.133 to 0.813] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.0582, Mixed Models Analysis; Mean Difference (Net) = 0.338, 95% CI 2-sided [-0.007 to 0.683] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.573, 95% CI 2-sided [0.232 to 0.914] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.0745, Mixed Models Analysis; Mean Difference (Net) = 0.324, 95% CI 2-sided [-0.020 to 0.668] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.043, 95% CI 2-sided [-0.337 to 0.422] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.9759, Mixed Models Analysis; Mean Difference (Net) = -0.116, 95% CI 2-sided [-0.501 to 0.268] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.7128, Mixed Models Analysis; Mean Difference (Net) = -0.186, 95% CI 2-sided [-0.565 to 0.192] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHPhe amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.6816, Mixed Models Analysis; Mean Difference (Net) = -0.195, 95% CI 2-sided [-0.582 to 0.192] — [estimate comment as in outcome 1, analysis 1]

34. Secondary Outcome: Summary of 1-OHPhe Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 1-OH-Phenanthrene (1-OHPhe) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.005 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | -2.014 (35.7667) | -30.659 (39.1914) | -21.599 (45.5212) | -47.691 (44.6728) | -54.224 (39.4318) | -56.563 (25.0593)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | -3.193 (33.2980) | -35.291 (32.2576) | -32.597 (38.1268) | -55.524 (30.9398) | -31.699 (156.6252) | -52.495 (28.1468)

35. Secondary Outcome: Summary of 1-OHP Amount Excreted and Absolute Change From Baseline (ug/24 Hour) by Study Group and Study Day (mITT Population)
Description: Summary of 1-hydroxypyrene (1-OHP) amount excreted (ug/24 hour) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.01 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/24 hour
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
ug/24 hour
  Day -1 | 0.463 (0.4552) | 0.446 (0.2545) | 0.592 (0.4884) | 0.688 (0.6987) | 0.473 (0.2597) | 0.446 (0.2616)
  Day 5 | 0.428 (0.2850) | 0.380 (0.2917) | 0.454 (0.2575) | 0.407 (0.3324) | 0.338 (0.2872) | 0.314 (0.2238)
  Day 7: number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Day 7 | 0.377 (0.1970) | 0.352 (0.2555) | 0.451 (0.3757) | 0.483 (0.4287) | 0.371 (0.3406) | 0.440 (0.4277)
  Change from Baseline (Day 5) | -0.034 (0.4123) | -0.066 (0.2799) | -0.138 (0.3833) | -0.281 (0.6769) | -0.135 (0.3196) | -0.132 (0.2950)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 40 | 41 | 25 | 25 | 27
  Change from Baseline (Day 7) | -0.085 (0.3795) | -0.077 (0.2851) | -0.141 (0.3754) | -0.213 (0.6848) | -0.094 (0.3427) | 0.010 (0.3450)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.948, 95% CI 2-sided [-1.146 to -0.750] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 1 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.019, 95% CI 2-sided [-1.242 to -0.796] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.172, 95% CI 2-sided [-1.358 to -0.986] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.196, 95% CI 2-sided [-1.409 to -0.983] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.049, 95% CI 2-sided [-1.239 to -0.859] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.200, 95% CI 2-sided [-1.414 to -0.986] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.337, 95% CI 2-sided [-1.574 to -1.099] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.345, 95% CI 2-sided [-1.616 to -1.075] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.452, 95% CI 2-sided [-1.685 to -1.219] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.339, 95% CI 2-sided [-1.608 to -1.071] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.348, 95% CI 2-sided [-1.577 to -1.118] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 6 is equal to zero on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.227, 95% CI 2-sided [-1.488 to -0.966] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.5646, Mixed Models Analysis; Mean Difference (Net) = -0.224, 95% CI 2-sided [-0.607 to 0.160] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.8765, Mixed Models Analysis; Mean Difference (Net) = -0.177, 95% CI 2-sided [-0.609 to 0.254] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.9954, Mixed Models Analysis; Mean Difference (Net) = -0.101, 95% CI 2-sided [-0.488 to 0.287] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.8665, Mixed Models Analysis; Mean Difference (Net) = -0.181, 95% CI 2-sided [-0.613 to 0.252] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.1165, Mixed Models Analysis; Mean Difference (Net) = -0.389, 95% CI 2-sided [-0.829 to 0.052] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.3896, Mixed Models Analysis; Mean Difference (Net) = -0.326, 95% CI 2-sided [-0.821 to 0.168] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0122, Mixed Models Analysis; Mean Difference (Net) = -0.504, 95% CI 2-sided [-0.934 to -0.074] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.3938, Mixed Models Analysis; Mean Difference (Net) = -0.320, 95% CI 2-sided [-0.807 to 0.167] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.8501, Mixed Models Analysis; Mean Difference (Net) = 0.176, 95% CI 2-sided [-0.237 to 0.589] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.031, 95% CI 2-sided [-0.435 to 0.496] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.2928, Mixed Models Analysis; Mean Difference (Net) = 0.299, 95% CI 2-sided [-0.117 to 0.715] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.027, 95% CI 2-sided [-0.439 to 0.493] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.011, 95% CI 2-sided [-0.453 to 0.475] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.9966, Mixed Models Analysis; Mean Difference (Net) = -0.118, 95% CI 2-sided [-0.640 to 0.403] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9976, Mixed Models Analysis; Mean Difference (Net) = -0.104, 95% CI 2-sided [-0.560 to 0.352] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: 1-OHP amount excreted (ug/24 hour) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.9976, Mixed Models Analysis; Mean Difference (Net) = -0.112, 95% CI 2-sided [-0.628 to 0.404] — [estimate comment as in outcome 1, analysis 1]

36. Secondary Outcome: Summary of 1-OHP Amount Excreted Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of 1-hydroxypyrene (1-OHP) amount excreted percent change from Baseline (%) is presented. Subjects with valid sample results are included. Original values reported as below the limit of quantitation (BLQ) were set to one-half of the LLOQ (0.01 ng/mL) for summarization and statistical analysis. Baseline = Day -1.
  24-hour urine collections occurred on Days -1, 5, and 7 beginning after the first morning void and any void prior to 07:00, and finished the following morning with the last void collected at approximately 07:00 (including first morning void).
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 27 | 28
percentage of change
  Day 5 | 14.604 (64.3632) | -9.171 (55.4282) | -3.632 (63.0769) | -22.640 (46.8991) | -19.442 (63.1149) | -9.058 (94.5456)
  Day 7 | 1.713 (40.2284) | -9.849 (58.6387) | -15.538 (49.5890) | -18.133 (51.8440) | -10.328 (72.1902) | 1.959 (68.3664)

37. Secondary Outcome: Summary of Urine Mutagenicity and Absolute Change From Baseline (Revertants/24 Hours) by Study Group and Study Day (mITT Population)
Description: Summary of urine mutagenicity (revertants/24 hours) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Baseline = Day -1.
  250 mL urine sample will be concentrated to 1 mL and used for urine mutagenicity testing. The measurement results will be reported as revertants/μL. The urine mutagenicity count in the 24 hour urine will be calculated as: Urine mutagenicity (revertants/24 hour) = Urine mutagenicity (revertants/250 mL) x urine volume/ urine sample volume in mL
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: revertants/24 hours
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 39 | 40 | 26 | 26 | 26
revertants/24 hours
  Day -1 | 42695.9 (31628.41) | 40627.1 (24929.42) | 31725.0 (22029.85) | 38042.0 (25874.21) | 39185.5 (23427.24) | 45475.7 (24556.04)
  Day 5: number analyzed (Participants) | 38 | 37 | 40 | 26 | 26 | 24
  Day 5 | 39814.0 (33030.58) | 21489.1 (15437.94) | 18917.1 (11973.55) | 3222.7 (4029.83) | 2450.8 (3355.41) | 3051.1 (3011.89)
  Day 7: number analyzed (Participants) | 38 | 37 | 40 | 25 | 24 | 24
  Day 7 | 40008.3 (32211.76) | 21884.6 (13846.21) | 23575.3 (16787.62) | 5231.0 (6316.63) | 2962.7 (4112.19) | 4642.7 (6147.86)
  Change from Baseline (Day 5): number analyzed (Participants) | 38 | 37 | 40 | 26 | 26 | 24
  Change from Baseline (Day 5) | -2881.9 (19517.06) | -20856.2 (22171.89) | -12807.9 (16642.34) | -34819.4 (24457.34) | -36734.7 (22541.48) | -41002.6 (24082.18)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 37 | 40 | 25 | 24 | 24
  Change from Baseline (Day 7) | -2687.6 (24781.58) | -17841.2 (21897.40) | -8149.7 (14961.88) | -33209.8 (25485.69) | -36626.8 (25513.32) | -42147.8 (23806.81)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 1 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 1 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 180.0, 95% CI 2-sided [164.9 to 195.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 1 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 1 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 181.1, 95% CI 2-sided [165.9 to 196.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 132.3, 95% CI 2-sided [117.2 to 147.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 137.3, 95% CI 2-sided [122.1 to 152.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 136.8, 95% CI 2-sided [122.0 to 151.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 150.8, 95% CI 2-sided [136.0 to 165.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 43.2, 95% CI 2-sided [25.1 to 61.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 61.7, 95% CI 2-sided [43.2 to 80.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 36.9, 95% CI 2-sided [18.6 to 55.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = 35.5, 95% CI 2-sided [16.7 to 54.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 6 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 6 is equal to zero on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 38.8, 95% CI 2-sided [19.9 to 57.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 6 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 6 is equal to zero on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 44.9, 95% CI 2-sided [26.0 to 63.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = -47.7, 95% CI 2-sided [-78.0 to -17.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0009, Mixed Models Analysis; Mean Difference (Net) = -43.8, 95% CI 2-sided [-74.1 to -13.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p = 0.0009, Mixed Models Analysis; Mean Difference (Net) = -43.2, 95% CI 2-sided [-73.2 to -13.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p = 0.0466, Mixed Models Analysis; Mean Difference (Net) = -30.2, 95% CI 2-sided [-60.2 to -0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -136.8, 95% CI 2-sided [-170.4 to -103.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -119.4, 95% CI 2-sided [-153.3 to -85.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -143.2, 95% CI 2-sided [-176.6 to -109.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -145.6, 95% CI 2-sided [-179.7 to -111.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 93.6, 95% CI 2-sided [60.0 to 127.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 92.4, 95% CI 2-sided [58.8 to 126.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 98.1, 95% CI 2-sided [64.6 to 131.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 106.0, 95% CI 2-sided [72.5 to 139.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 4.5, 95% CI 2-sided [-32.0 to 40.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.7714, Mixed Models Analysis; Mean Difference (Net) = 16.8, 95% CI 2-sided [-20.0 to 53.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = -1.9, 95% CI 2-sided [-38.3 to 34.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: Urine Mutagenicity (revertants/24 hours) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 0.9926, Mixed Models Analysis; Mean Difference (Net) = -9.4, 95% CI 2-sided [-46.4 to 27.6] — [estimate comment as in outcome 1, analysis 1]

38. Secondary Outcome: Summary of Urine Mutagenicity Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of urine mutagenicity percent change from Baseline (%) by study group and study day is presented. Baseline = Day -1.
  250 mL urine sample will be concentrated to 1 mL and used for urine mutagenicity testing. The measurement results will be reported as revertants/μL. The urine mutagenicity count in the 24 hour urine will be calculated as: Urine mutagenicity (revertants/24 hour) = Urine mutagenicity (revertants/250 mL) x urine volume/ urine sample volume in mL
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 37 | 40 | 26 | 26 | 23
percentage of change
  Day 5 | 6.059 (60.6504) | -40.200 (37.5319) | -27.954 (45.8289) | -91.239 (9.0409) | -93.056 (7.6922) | -91.057 (9.3363)
  Day 7: number analyzed (Participants) | 38 | 37 | 40 | 25 | 24 | 23
  Day 7 | 7.844 (62.4696) | -26.765 (75.6831) | -14.729 (60.1017) | -84.415 (16.2799) | -87.632 (25.0981) | -88.904 (11.3419)

39. Secondary Outcome: Summary of Whole Blood COHb and Absolute Change From Baseline (% Saturation) by Study Group and Study Day (mITT Population)
Description: Summary of whole blood carboxyhemoglobin [COHb] (% saturation) by study group on Days -1, 5 and 7, and absolute change from Baseline on Days 5 and 7 are presented. Subjects with valid sample results are included. Baseline = Day -1.
  The blood sample for COHb was collected approximately 21:30 on Days -1, 5, and 7 after subjects abstained from product use, as appropriate, for at least 15 minutes prior to blood draw for COHb.
  Absolute change from baseline was calculated as: Post Randomization Value - Baseline Value
Time Frame: Baseline (Day -1), Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % Saturation
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 28 | 28
% Saturation
  Day -1 | 6.68 (1.815) | 6.81 (1.650) | 7.11 (1.927) | 7.23 (2.269) | 6.98 (1.711) | 6.89 (2.038)
  Day 5 | 6.53 (1.599) | 4.50 (1.216) | 4.91 (1.304) | 1.78 (0.169) | 1.73 (0.272) | 1.79 (0.281)
  Day 7: number analyzed (Participants) | 38 | 42 | 40 | 25 | 26 | 27
  Day 7 | 6.77 (1.516) | 4.61 (1.244) | 5.11 (1.274) | 1.85 (0.302) | 1.82 (0.388) | 1.79 (0.281)
  Change from Baseline (Day 5) | -0.15 (1.231) | -2.32 (1.328) | -2.20 (1.251) | -5.45 (2.253) | -5.25 (1.711) | -5.10 (1.903)
  Change from Baseline (Day 7): number analyzed (Participants) | 38 | 42 | 40 | 25 | 26 | 27
  Change from Baseline (Day 7) | 0.09 (1.394) | -2.20 (1.304) | -1.98 (1.193) | -5.28 (2.269) | -5.22 (1.684) | -5.04 (1.893)
Statistical Analysis 1: Comparison: GROUP 1: Continue Smoking; Null hypothesis: Whole Blood COHB (% Saturation) in Group 1 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 1 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 1 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 1 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.872, 95% CI 2-sided [1.810 to 1.935] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: GROUP 1: Continue Smoking; Null hypothesis: Whole Blood COHB (% Saturation) in Group 1 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 1 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 1 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 1 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.913, 95% CI 2-sided [1.851 to 1.976] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.467, 95% CI 2-sided [1.408 to 1.525] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GROUP 2: OTDN Product 1; Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.493, 95% CI 2-sided [1.434 to 1.551] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.550, 95% CI 2-sided [1.490 to 1.609] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: GROUP 3: OTDN Product 2; Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.594, 95% CI 2-sided [1.533 to 1.654] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.557, 95% CI 2-sided [0.482 to 0.631] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GROUP 4: OTDN Product 1; Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.589, 95% CI 2-sided [0.514 to 0.665] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.533, 95% CI 2-sided [0.461 to 0.605] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GROUP 5: OTDN Product 2; Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.588, 95% CI 2-sided [0.514 to 0.662] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: Whole Blood COHB (% Saturation) in Group 6 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 6 is NOT equal to zero on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 6 is equal to zero on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 6 is NOT equal to zero on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.580, 95% CI 2-sided [0.508 to 0.652] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: GROUP 6: Tobacco Cessation; Null hypothesis: Whole Blood COHB (% Saturation) in Group 6 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 6 is NOT equal to zero on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 6 is equal to zero on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 6 is NOT equal to zero on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.580, 95% CI 2-sided [0.507 to 0.653] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to Group 1 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.406, 95% CI 2-sided [-0.526 to -0.285] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: GROUP 1: Continue Smoking vs GROUP 2: OTDN Product 1; Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to Group 1 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.421, 95% CI 2-sided [-0.541 to -0.300] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to Group 1 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.323, 95% CI 2-sided [-0.444 to -0.201] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: GROUP 1: Continue Smoking vs GROUP 3: OTDN Product 2; Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to Group 1 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.320, 95% CI 2-sided [-0.442 to -0.198] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to Group 1 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.315, 95% CI 2-sided [-1.453 to -1.178] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: GROUP 1: Continue Smoking vs GROUP 4: OTDN Product 1; Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to Group 1 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.324, 95% CI 2-sided [-1.463 to -1.186] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to Group 1 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to Group 1 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.339, 95% CI 2-sided [-1.473 to -1.205] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: GROUP 1: Continue Smoking vs GROUP 5: OTDN Product 2; Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to Group 1 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to Group 1 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.325, 95% CI 2-sided [-1.461 to -1.190] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to Group 6 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.887, 95% CI 2-sided [0.757 to 1.016] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: GROUP 2: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 2 is equal to Group 6 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 2 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.912, 95% CI 2-sided [0.782 to 1.043] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to Group 6 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to Group 6 on Day 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.970, 95% CI 2-sided [0.839 to 1.100] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: GROUP 3: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 3 is equal to Group 6 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 3 is NOT equal to Group 6 on Day 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.013, 95% CI 2-sided [0.882 to 1.145] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to Group 6 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9999, Mixed Models Analysis; Mean Difference (Net) = -0.023, 95% CI 2-sided [-0.168 to 0.122] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: GROUP 4: OTDN Product 1 vs GROUP 6: Tobacco Cessation; Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 4 is equal to Group 6 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 4 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.009, 95% CI 2-sided [-0.138 to 0.155] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to Group 6 on Day 5. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to Group 6 on Day 5. (mITT Population); p = 0.9577, Mixed Models Analysis; Mean Difference (Net) = -0.047, 95% CI 2-sided [-0.189 to 0.095] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: GROUP 5: OTDN Product 2 vs GROUP 6: Tobacco Cessation; Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood COHB (% Saturation) in Group 5 is equal to Group 6 on Day 7. Alternate hypothesis: Whole Blood COHB (% Saturation) in Group 5 is NOT equal to Group 6 on Day 7. (mITT Population); p = 1.0000, Mixed Models Analysis; Mean Difference (Net) = 0.008, 95% CI 2-sided [-0.136 to 0.152] — [estimate comment as in outcome 1, analysis 1]

40. Secondary Outcome: Summary of Whole Blood COHb Percent Change From Baseline (%) by Study Group and Study Day (mITT Population)
Description: Summary of whole blood carboxyhemoglobin (COHb) percent change from Baseline (%) is presented. Subjects with valid sample results are included. Baseline = Day -1.
  The blood sample for COHb was collected approximately 21:30 on Days -1, 5, and 7 after subjects abstained from product use, as appropriate, for at least 15 minutes prior to blood draw for COHb.
  % change from Baseline = (Post Randomization Value - Baseline Value) / Baseline Value x 100 %
Time Frame: Day 5 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 28 | 28
percentage of change
  Day 5 | 0.459 (19.3191) | -32.762 (15.6487) | -29.807 (11.1205) | -73.352 (7.5619) | -73.827 (7.7024) | -72.424 (7.7658)
  Day 7: number analyzed (Participants) | 38 | 42 | 40 | 25 | 26 | 27
  Day 7 | 5.451 (25.3747) | -31.264 (14.3934) | -26.160 (14.0914) | -71.853 (10.0793) | -72.896 (7.7120) | -72.391 (6.4588)

41. Secondary Outcome: Cigarette Consumption by Study Group and Study Day (mITT Population)
Description: Summary of cigarette consumption, as number of cigarettes smoked per day (CPD), by study group and study day is presented. Baseline = Average of Days -2 and -1.
Time Frame: Day -1 and Day -2 (Baseline), Day 1, Day 2, Day 3, Day 4, Day 5, Day 6 and Day 7
Population: Modified ITT: All randomized subjects who used at least one study product after randomization (except Group 6) and had a valid baseline and at least one post-baseline biomarker measure.
  Subjects in Groups 4, 5, and 6 were instructed to refrain from smoking cigarettes after Day -1 in compliance with the product use group assignment. No CPD data was collected for these groups on Days 1 through 7 and the Number of Participants Analyzed is reported as '0' in the data table.
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
Number analyzed (Participants) | 38 | 42 | 41 | 26 | 28 | 28
cigarettes per day
  Day -2 | 16.6 (3.80) | 16.7 (4.15) | 17.8 (4.82) | 16.7 (4.95) | 16.8 (5.08) | 16.2 (3.68)
  Day -1 | 17.4 (4.52) | 17.6 (4.52) | 18.8 (6.17) | 17.3 (4.67) | 17.0 (4.73) | 17.5 (4.20)
  Baseline | 17.00 (3.958) | 17.17 (4.131) | 18.33 (5.197) | 17.02 (4.568) | 16.89 (4.661) | 16.82 (3.735)
  Day 1: number analyzed (Participants) | 38 | 42 | 41 | 0 | 0 | 0
  Day 1 | 16.4 (3.71) | 8.1 (2.14) | 8.8 (2.51) |  |  |
  Day 2: number analyzed (Participants) | 38 | 42 | 41 | 0 | 0 | 0
  Day 2 | 16.0 (3.70) | 8.2 (2.35) | 8.7 (2.54) |  |  |
  Day 3: number analyzed (Participants) | 38 | 41 | 41 | 0 | 0 | 0
  Day 3 | 15.7 (4.51) | 8.2 (2.09) | 8.8 (2.54) |  |  |
  Day 4: number analyzed (Participants) | 38 | 41 | 41 | 0 | 0 | 0
  Day 4 | 15.7 (3.88) | 8.1 (2.20) | 8.7 (2.53) |  |  |
  Day 5: number analyzed (Participants) | 38 | 41 | 41 | 0 | 0 | 0
  Day 5 | 16.1 (4.51) | 8.2 (2.27) | 8.6 (2.61) |  |  |
  Day 6: number analyzed (Participants) | 38 | 41 | 41 | 0 | 0 | 0
  Day 6 | 15.5 (4.00) | 8.2 (2.14) | 8.7 (2.58) |  |  |
  Day 7: number analyzed (Participants) | 38 | 41 | 41 | 0 | 0 | 0
  Day 7 | 17.1 (4.43) | 8.2 (2.10) | 8.8 (2.67) |  |  |

42. Secondary Outcome: Summary of VERVE® Product Usage by Study Group and Study Day (mITT Population)
Description: Summary of VERVE® Product Used Per Day by Study Group and Study Day is presented. Only study groups that received the test product (VERVE® Discs or VERVE® Chews) are shown. Results are stratified by product flavor (Green Mint, Blue Mint and overall).
Time Frame: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: products per day
Groups:
- GROUP 2: OTDN Product 1 (VERVE® Green Mint Discs): Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 product units per day for 7 days.
  OTDN product 1: Oral tobacco-derived nicotine product (VERVE® Green Mint Discs)
- GROUP 2: OTDN Product 1 (VERVE® Blue Mint Discs): Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 product units per day for 7 days.
  OTDN product 1: Oral tobacco-derived nicotine product (VERVE® Blue Mint Discs)
- GROUP 2: OTDN Product 1 (VERVE® Discs Total): Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 product units per day for 7 days.
  OTDN product 1: Oral tobacco-derived nicotine product (VERVE® Discs Total)
- GROUP 3: OTDN Product 2 (VERVE® Green Mint Chews): Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 product units per day for 7 days.
  OTDN product 2: Oral tobacco-derived nicotine product (VERVE® Green Mint Chews)
- GROUP 3: OTDN Product 2 (VERVE® Blue Mint Chews): Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 product units per day for 7 days.
  OTDN product 2: Oral tobacco-derived nicotine product (VERVE® Blue Mint Chews)
- GROUP 3: OTDN Product 2 (VERVE® Chews Total): Subjects will reduce their normal daily cigarette consumption by at least 50% of their baseline CPD and use at least 3 product units per day for 7 days.
  OTDN product 2: Oral tobacco-derived nicotine product (VERVE® Chews Total)
- GROUP 4: OTDN Product 1 (VERVE® Green Mint Discs): Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine product, using at least 3 product units per day for 7 days.
  OTDN product 1: Oral tobacco-derived nicotine product (VERVE® Green Mint Discs)
- GROUP 4: OTDN Product 1 (VERVE® Blue Mint Discs): Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine product, using at least 3 product units per day for 7 days.
  OTDN product 1: Oral tobacco-derived nicotine product (VERVE® Blue Mint Discs)
- GROUP 4: OTDN Product 1 (VERVE® Discs Total): Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine product, using at least 3 product units per day for 7 days.
  OTDN product 1: Oral tobacco-derived nicotine product (VERVE® Discs Total)
- GROUP 5: OTDN Product 2 (VERVE® Green Mint Chews): Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine product, using at least 3 product units per day for 7 days.
  OTDN product 2: Oral tobacco-derived nicotine product (VERVE® Green Mint Chews)
- GROUP 5: OTDN Product 2 (VERVE® Blue Mint Chews): Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine product, using at least 3 product units per day for 7 days.
  OTDN product 2: Oral tobacco-derived nicotine product (VERVE® Blue Mint Chews)
- GROUP 5: OTDN Product 2 (VERVE® Chews Total): Subjects will completely switch to exclusive use of an oral tobacco-derived nicotine product, using at least 3 product units per day for 7 days.
  OTDN product 2: Oral tobacco-derived nicotine product (VERVE® Chews Total)
Arm/Group | GROUP 2: OTDN Product 1 (VERVE® Green Mint Discs) | GROUP 2: OTDN Product 1 (VERVE® Blue Mint Discs) | GROUP 2: OTDN Product 1 (VERVE® Discs Total) | GROUP 3: OTDN Product 2 (VERVE® Green Mint Chews) | GROUP 3: OTDN Product 2 (VERVE® Blue Mint Chews) | GROUP 3: OTDN Product 2 (VERVE® Chews Total) | GROUP 4: OTDN Product 1 (VERVE® Green Mint Discs) | GROUP 4: OTDN Product 1 (VERVE® Blue Mint Discs) | GROUP 4: OTDN Product 1 (VERVE® Discs Total) | GROUP 5: OTDN Product 2 (VERVE® Green Mint Chews) | GROUP 5: OTDN Product 2 (VERVE® Blue Mint Chews) | GROUP 5: OTDN Product 2 (VERVE® Chews Total)
Number analyzed (Participants) | 42 | 42 | 42 | 41 | 41 | 41 | 26 | 26 | 26 | 28 | 28 | 28
products per day
  Day 1: number analyzed (Participants) | 35 | 33 | 42 | 37 | 31 | 41 | 25 | 16 | 26 | 26 | 16 | 28
  Day 1 | 4.2 (2.41) | 3.5 (2.73) | 6.3 (3.74) | 3.9 (2.31) | 3.0 (1.74) | 5.8 (2.78) | 8.9 (6.29) | 4.8 (6.41) | 11.5 (8.87) | 9.0 (5.88) | 4.5 (3.79) | 10.9 (7.38)
  Day 2: number analyzed (Participants) | 37 | 33 | 42 | 35 | 27 | 40 | 25 | 14 | 26 | 26 | 13 | 28
  Day 2 | 3.6 (2.02) | 4.2 (2.17) | 6.5 (2.96) | 3.3 (1.95) | 3.4 (1.42) | 5.2 (2.36) | 8.2 (6.37) | 6.9 (8.76) | 11.6 (8.60) | 7.7 (5.35) | 6.9 (4.87) | 10.4 (7.71)
  Day 3: number analyzed (Participants) | 34 | 33 | 42 | 35 | 30 | 41 | 24 | 13 | 26 | 24 | 15 | 28
  Day 3 | 3.9 (2.05) | 3.7 (1.76) | 6.0 (2.77) | 3.6 (2.13) | 3.5 (1.38) | 5.6 (2.76) | 7.8 (5.64) | 7.7 (9.61) | 11.0 (9.61) | 8.2 (5.75) | 6.0 (4.46) | 10.2 (7.03)
  Day 4: number analyzed (Participants) | 30 | 35 | 42 | 32 | 29 | 41 | 23 | 9 | 25 | 25 | 15 | 28
  Day 4 | 3.9 (2.35) | 3.6 (2.32) | 5.8 (3.14) | 3.7 (2.76) | 3.9 (2.08) | 5.6 (3.15) | 8.3 (6.98) | 8.7 (8.70) | 10.8 (9.22) | 7.0 (4.73) | 6.5 (4.79) | 9.7 (6.93)
  Day 5: number analyzed (Participants) | 32 | 32 | 41 | 36 | 31 | 41 | 23 | 11 | 26 | 23 | 15 | 28
  Day 5 | 3.3 (2.10) | 3.6 (1.72) | 5.4 (2.34) | 3.5 (1.87) | 3.5 (1.67) | 5.7 (2.82) | 7.9 (7.15) | 10.7 (10.26) | 11.5 (11.13) | 7.1 (5.17) | 6.5 (4.84) | 9.4 (7.33)
  Day 6: number analyzed (Participants) | 31 | 33 | 42 | 30 | 30 | 40 | 25 | 9 | 26 | 25 | 14 | 28
  Day 6 | 4.0 (2.30) | 3.6 (2.30) | 5.8 (2.73) | 3.9 (2.78) | 4.4 (2.75) | 6.2 (4.50) | 6.9 (5.89) | 9.9 (9.83) | 10.1 (9.42) | 6.0 (4.31) | 6.2 (5.10) | 8.5 (5.92)
  Day 7: number analyzed (Participants) | 28 | 31 | 42 | 27 | 28 | 41 | 21 | 12 | 24 | 23 | 14 | 26
  Day 7 | 3.8 (1.99) | 4.0 (2.44) | 5.4 (3.04) | 4.4 (2.38) | 4.6 (2.99) | 6.1 (4.81) | 8.1 (5.41) | 6.2 (3.93) | 10.2 (7.00) | 6.7 (4.99) | 5.3 (4.65) | 8.8 (6.08)

43. Secondary Outcome: Summary of VERVE® Product Use Duration by Study Group and Study Day (mITT Population)
Description: Summary of average VERVE® product use duration (minutes) by Study Group and Study Day is presented. Only study groups that received the test product (VERVE® Discs or VERVE® Chews) are shown. Results are stratified by product flavor (Green Mint, Blue Mint and overall).
Time Frame: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | GROUP 2: OTDN Product 1 (VERVE® Green Mint Discs) | GROUP 2: OTDN Product 1 (VERVE® Blue Mint Discs) | GROUP 2: OTDN Product 1 (VERVE® Discs Total) | GROUP 3: OTDN Product 2 (VERVE® Green Mint Chews) | GROUP 3: OTDN Product 2 (VERVE® Blue Mint Chews) | GROUP 3: OTDN Product 2 (VERVE® Chews Total) | GROUP 4: OTDN Product 1 (VERVE® Green Mint Discs) | GROUP 4: OTDN Product 1 (VERVE® Blue Mint Discs) | GROUP 4: OTDN Product 1 (VERVE® Discs Total) | GROUP 5: OTDN Product 2 (VERVE® Green Mint Chews) | GROUP 5: OTDN Product 2 (VERVE® Blue Mint Chews) | GROUP 5: OTDN Product 2 (VERVE® Chews Total)
Number analyzed (Participants) | 42 | 42 | 42 | 41 | 41 | 41 | 26 | 26 | 26 | 28 | 28 | 28
minutes
  Day 1: number analyzed (Participants) | 35 | 33 | 42 | 36 | 31 | 41 | 25 | 16 | 26 | 26 | 16 | 28
  Day 1 | 16.91 (9.058) | 19.06 (7.981) | 17.37 (7.486) | 16.81 (7.429) | 15.40 (4.389) | 16.38 (6.312) | 21.04 (12.430) | 36.07 (60.238) | 24.49 (20.627) | 24.03 (13.900) | 28.80 (29.840) | 23.40 (14.369)
  Day 2: number analyzed (Participants) | 37 | 33 | 42 | 35 | 27 | 40 | 25 | 14 | 26 | 26 | 13 | 28
  Day 2 | 17.77 (12.379) | 20.10 (10.256) | 18.03 (8.374) | 16.17 (8.430) | 15.46 (4.755) | 16.41 (7.557) | 19.75 (12.736) | 24.28 (18.445) | 20.67 (13.519) | 23.75 (16.970) | 23.98 (16.273) | 23.31 (15.503)
  Day 3: number analyzed (Participants) | 34 | 33 | 42 | 35 | 30 | 41 | 24 | 13 | 26 | 24 | 15 | 28
  Day 3 | 17.83 (11.425) | 19.40 (13.169) | 18.43 (11.026) | 17.52 (10.282) | 18.10 (7.953) | 17.66 (8.972) | 22.19 (14.651) | 17.35 (10.420) | 21.50 (14.545) | 24.37 (16.063) | 23.20 (17.406) | 23.92 (15.846)
  Day 4: number analyzed (Participants) | 30 | 35 | 42 | 32 | 29 | 41 | 23 | 9 | 25 | 25 | 15 | 28
  Day 4 | 15.78 (7.870) | 19.65 (9.810) | 16.73 (7.420) | 18.63 (14.374) | 15.56 (5.719) | 17.42 (11.163) | 23.67 (16.357) | 18.55 (11.495) | 23.33 (15.876) | 27.80 (22.588) | 33.71 (35.998) | 26.30 (22.554)
  Day 5: number analyzed (Participants) | 32 | 32 | 41 | 36 | 31 | 41 | 23 | 11 | 26 | 23 | 15 | 28
  Day 5 | 21.38 (13.978) | 23.22 (14.124) | 20.20 (11.398) | 17.67 (10.156) | 16.96 (8.840) | 17.48 (10.334) | 22.81 (17.683) | 21.08 (14.347) | 21.76 (17.151) | 25.71 (20.315) | 35.75 (34.492) | 29.26 (28.160)
  Day 6: number analyzed (Participants) | 31 | 33 | 42 | 30 | 30 | 40 | 25 | 9 | 26 | 25 | 14 | 28
  Day 6 | 17.87 (11.063) | 23.23 (14.472) | 18.77 (9.691) | 16.45 (8.468) | 16.94 (5.422) | 16.77 (6.913) | 24.05 (19.149) | 17.98 (12.472) | 23.86 (18.887) | 28.84 (24.557) | 30.48 (23.753) | 27.44 (22.541)
  Day 7: number analyzed (Participants) | 28 | 30 | 42 | 27 | 28 | 41 | 21 | 11 | 24 | 23 | 14 | 26
  Day 7 | 20.48 (21.835) | 23.28 (14.382) | 19.92 (12.807) | 17.48 (11.218) | 18.20 (11.249) | 16.31 (8.677) | 25.74 (18.642) | 16.95 (10.356) | 23.94 (17.928) | 29.14 (24.030) | 33.44 (24.807) | 28.08 (23.037)

44. Secondary Outcome: Summary of Total Duration (Min) of VERVE® Product Per Day by Study Group and Study Day (mITT Population)
Description: Summary of total duration (minutes) of VERVE® product per day by Study Group and Study Day. Only study groups that received the test product (VERVE® Discs or VERVE® Chews) are shown. Results are stratified by product flavor (Green Mint, Blue Mint and overall).
Time Frame: Day 1, Day 2, Day 3, Day 4, Day 5, Day 6 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | GROUP 2: OTDN Product 1 (VERVE® Green Mint Discs) | GROUP 2: OTDN Product 1 (VERVE® Blue Mint Discs) | GROUP 2: OTDN Product 1 (VERVE® Discs Total) | GROUP 3: OTDN Product 2 (VERVE® Green Mint Chews) | GROUP 3: OTDN Product 2 (VERVE® Blue Mint Chews) | GROUP 3: OTDN Product 2 (VERVE® Chews Total) | GROUP 4: OTDN Product 1 (VERVE® Green Mint Discs) | GROUP 4: OTDN Product 1 (VERVE® Blue Mint Discs) | GROUP 4: OTDN Product 1 (VERVE® Discs Total) | GROUP 5: OTDN Product 2 (VERVE® Green Mint Chews) | GROUP 5: OTDN Product 2 (VERVE® Blue Mint Chews) | GROUP 5: OTDN Product 2 (VERVE® Chews Total)
Number analyzed (Participants) | 42 | 42 | 42 | 41 | 41 | 41 | 26 | 26 | 26 | 28 | 28 | 28
minutes
  Day 1: number analyzed (Participants) | 35 | 33 | 42 | 36 | 31 | 41 | 25 | 16 | 26 | 26 | 16 | 28
  Day 1 | 66.6 (60.86) | 53.3 (35.94) | 96.4 (73.30) | 62.8 (57.27) | 43.3 (28.82) | 87.0 (59.79) | 157.8 (128.82) | 68.2 (69.75) | 181.8 (124.40) | 176.2 (140.91) | 66.8 (52.65) | 190.0 (150.02)
  Day 2: number analyzed (Participants) | 37 | 33 | 42 | 35 | 27 | 40 | 25 | 14 | 26 | 26 | 13 | 28
  Day 2 | 55.4 (43.38) | 75.0 (65.29) | 106.1 (93.40) | 54.4 (64.55) | 45.0 (20.73) | 75.8 (59.77) | 136.1 (123.65) | 106.6 (127.33) | 167.1 (133.55) | 158.1 (143.12) | 127.4 (134.79) | 180.0 (157.77)
  Day 3: number analyzed (Participants) | 34 | 33 | 42 | 35 | 30 | 41 | 24 | 13 | 26 | 24 | 15 | 28
  Day 3 | 58.9 (45.94) | 70.4 (77.83) | 95.8 (85.57) | 55.8 (47.73) | 53.7 (28.27) | 81.2 (57.39) | 143.3 (155.53) | 94.8 (124.33) | 165.8 (157.13) | 168.0 (158.06) | 112.3 (118.36) | 183.9 (161.66)
  Day 4: number analyzed (Participants) | 30 | 35 | 42 | 32 | 29 | 41 | 23 | 9 | 25 | 25 | 15 | 28
  Day 4 | 53.3 (50.87) | 56.4 (50.96) | 78.7 (60.02) | 59.2 (65.29) | 51.8 (36.46) | 76.1 (62.69) | 147.1 (151.60) | 107.4 (107.71) | 160.0 (146.22) | 160.5 (169.97) | 143.5 (144.53) | 193.0 (192.40)
  Day 5: number analyzed (Participants) | 32 | 32 | 41 | 36 | 31 | 41 | 23 | 11 | 26 | 23 | 15 | 28
  Day 5 | 55.5 (40.23) | 70.5 (71.71) | 87.8 (76.80) | 52.0 (51.65) | 52.9 (48.87) | 74.8 (58.45) | 143.7 (160.99) | 122.5 (96.15) | 160.9 (163.65) | 154.5 (159.58) | 161.8 (174.46) | 191.8 (185.32)
  Day 6: number analyzed (Participants) | 31 | 33 | 42 | 30 | 30 | 40 | 25 | 9 | 26 | 25 | 14 | 28
  Day 6 | 51.9 (32.63) | 62.2 (55.51) | 82.7 (58.15) | 57.4 (56.87) | 60.3 (50.07) | 74.8 (60.34) | 148.0 (182.96) | 114.1 (115.23) | 166.3 (176.75) | 157.0 (183.23) | 173.3 (213.39) | 191.0 (206.39)
  Day 7: number analyzed (Participants) | 28 | 30 | 42 | 27 | 28 | 41 | 21 | 11 | 24 | 23 | 14 | 26
  Day 7 | 55.2 (40.88) | 75.7 (62.68) | 82.5 (63.51) | 60.9 (46.53) | 73.8 (71.37) | 76.3 (77.57) | 164.3 (170.36) | 92.2 (121.70) | 167.4 (164.72) | 154.0 (173.42) | 136.8 (132.81) | 182.8 (178.99)

45. Secondary Outcome: Summary of Response for Willingness to Use Cigarettes Again Bipolar VAS Scores for Cigarettes by Category, Study Group and Study Product (mITT Population)
Description: Summary of subject responses to "Use the Product (Cigarette) Again" Bipolar Visual Analogue Scale (VAS) Scores for cigarettes is presented. The Use the Product Again Bipolar VAS is a 100 mm scale ranging from 0 mm ("Definitely Would Not") to 100 mm ("Definitely Would"). The bipolar score is calculated by subtracting 50 from the original VAS score, then categorizing into three categories: -50 to <0, 0, and >0 to 50. Higher scores are associated with greater willingness to use the cigarettes again. Mean and standard deviation of the bipolar VAS score per category is shown.
  The "Use the Product Again" VAS Score was given to subjects on Day 7 at 21:30 (±30 minutes) during the product use period.
  The data shown are the means calculated from only those participants with scores in the corresponding category ('-50 to <0', '0' and '>0 to 50').
Time Frame: Data collected on Day 7 at 21:30 (±30 minutes) during the product use period
Population: The mITT population consisted of all randomized subjects who used at least one study product after randomization (except Group 6) and had a valid baseline and at least one post-baseline biomarker measure. Only subjects who were smoked their own cigarette brand were asked to complete the "Use Product (Cigarette) Again" VAS score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2
Number analyzed (Participants) | 38 | 42 | 39
units on a scale
  -50 to <0: number analyzed (Participants) | 1 | 7 | 6
  -50 to <0 | -3.0 | -20.7 (18.14) | -17.0 (15.80)
  0: number analyzed (Participants) | 1 | 1 | 0
  0 | 0.0 | 0.0 |
  >0 to 50: number analyzed (Participants) | 36 | 34 | 33
  >0 to 50 | 37.3 (14.67) | 37.1 (14.92) | 30.8 (16.13)

46. Secondary Outcome: Summary of Response for Willingness to Use the VERVE® Product Again Bipolar VAS Scores for Cigarettes by Category, Study Group and Study Product (mITT Population)
Description: Summary of subject responses to "Use the Product (VERVE®) Again" Bipolar Visual Analogue Scale (VAS) Scores for the VERVE® test products are presented. The Use the Product Again Bipolar VAS is a 100 mm scale ranging from 0 mm ("Definitely Would Not") to 100 mm ("Definitely Would"). The bipolar score is calculated by subtracting 50 from the original VAS score, then categorizing into three categories: -50 to <0, 0, and >0 to 50. Higher scores are associated with greater willingness to use the VERVE® product again. Mean and standard deviation of the bipolar VAS score per category is shown.
  The "Use the Product Again" VAS Score was given to subjects on Day 7 at 21:30 (±30 minutes) during the product use period.
  The data shown are the means calculated from only those participants with scores in the corresponding category ('-50 to <0', '0' and '>0 to 50').
Time Frame: Data collected on Day 7 at 21:30 (±30 minutes) during the product use period
Population: The mITT population consisted of all randomized subjects who used at least one study product after randomization (except Group 6) and had a valid baseline and at least one post-baseline biomarker measure. Only subjects who used the VERVE® product were asked to complete the "Use Product (VERVE®) Again" VAS score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2
Number analyzed (Participants) | 42 | 40 | 25 | 25
units on a scale
  -50 to <0: number analyzed (Participants) | 14 | 13 | 14 | 8
  -50 to <0 | -36.5 (18.92) | -27.1 (19.59) | -30.7 (19.11) | -27.3 (15.70)
  0: number analyzed (Participants) | 3 | 2 | 0 | 1
  0 | 0.0 (0.00) | 0.0 (0.00) |  | 0.0
  >0 to 50: number analyzed (Participants) | 25 | 25 | 11 | 16
  >0 to 50 | 25.4 (14.02) | 29.1 (13.02) | 27.6 (17.19) | 31.0 (15.59)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from subjects' first study product use [VERVE® product trial on Day -3] through discharge on Day 8 or Early Termination for a total of up to 11 days.
Description: The Safety Population includes all subjects who tried the test product at least once during the study, including those subjects who participated only in the product trial phase. AEs will be monitored and recorded from the time of the first product use (VERVE® product trial at Check-in on Day -3) through the End-of-Study (or Early Termination). Events captured between Screening and the first study product use will be documented as baseline signs and symptoms (in medical history) and not AEs.
Arm/Group | Product Trial | GROUP 1: Continue Smoking | GROUP 2: OTDN Product 1 | GROUP 3: OTDN Product 2 | GROUP 4: OTDN Product 1 | GROUP 5: OTDN Product 2 | GROUP 6: Tobacco Cessation
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/40 | 0/42 | 0/41 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/40 | 0/42 | 0/41 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 66/231 | 6/40 | 12/42 | 14/41 | 14/30 | 14/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Product Trial (N=231) | GROUP 1: Continue Smoking (N=40) | GROUP 2: OTDN Product 1 (N=42) | GROUP 3: OTDN Product 2 (N=41) | GROUP 4: OTDN Product 1 (N=30) | GROUP 5: OTDN Product 2 (N=30) | GROUP 6: Tobacco Cessation (N=30)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 4 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sputum abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 45 (47) | 3 (3) | 3 (3) | 5 (5) | 4 (4) | 2 (2) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: ALCS-RDS-18-04-VRV Protocol Version 1 (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT03692078/Prot_000.pdf
  • Study Protocol: ALCS-RDS-18-04-VRV Protocol Version 2 (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT03692078/Prot_001.pdf
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03692078/SAP_002.pdf